

### CLINICAL STUDY REPORT WIL-30

### 16.1.9 Documentation of Statistical Methods



### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30

Date of Issue: 2017-04-26

Version Number: 1.0


| Sponsor: | Octapharma AG |
|---|---|
| Title of Protocol: | Clinical Study to Investigate the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of <i>Wilate</i> in Previously Treated Pediatric Patients with Severe Hemophilia A |
| Protocol Version/Date: | Version 1.0 / 2017-04-26 |
| CRF Version: | TBD |
| Supersedes SAP Version: | None |


This document contains confidential information which must not be disclosed to anyone other than the involved CRO. This information should not be used for any purpose other than the evaluation of the clinical investigation without prior written consent of Octapharma.

No part of this document may be reproduced or stored in a retrieval system or transmitted in any other form or by any other means.



### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30


Date of Issue: 2017-04-26


### **Document authorization**





# STATISTICAL ANALYSIS PLAN ProtocolNo:WIL-30 Version Number: 1.0 Date of Issue: 2017-04-26 

### Consistency check with the Protocol (one option to be selected)

| X | This is to confirm that as part of the SAP finalization consistency check with the curren protocol / protocol amendment was performed by the trial statistician, and no changes to the protocol (statistical section) are required |
|---|---|
| | Changes to the analysis principles were required, and the responsible team has confirmed commitment to update the study protocol |
| | Changes to the analysis principles were required (as outlined in revision history section of this SAP), however it was not feasible to update the study protocol, for the reason |





| STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 | |
|-----------------------------------------------|--------------|
| Version Number: 1.0 | D 4 - 6 27 |
| Date of Issue: 2017-04-26 | |

### Change control

| Date | Author | Reason | Version |
|------------|--------|--------|---------|
| 2017-04-26 | | | 1.0 |



Protocol No: WIL-30


Date of Issue: 2017-04-26


### TABLE OF CONTENTS

| Document authorization | |
|---|---|
| Consistency check with the Protocol (one option to be selected) | 3 |
| Change control | |
| Table of contents | |
| List of abbreviations | |
| 1 Study material | |
| 2 Study information | |
| 2.1 Primary objective | |
| 2.2 Secondary objective | |
| 2.3 Additional Objective: | |
| 2.4 Study design | |
| 2.5 Planned sample size | |
| 3 General Information | |
| 3.1 Background details | |
| 3.2 Deviations from the trial protocol with regard to statistical analyses | |
| 3.3 Individual protocol deviations | |
| 4 Analysis Populations | |
| 4.1 Safety set | |
| 4.2 Full analysis set | |
| 4.3 Pharmacokinetic set | |
| 4.4 Per-protocol set | |
| 4.5 Surgery set | |
| 4.6 Subgroup analyses | |
| 5 Statistical Analyses | |
| 5.1 Conventions | |
| 5.1.1 Baseline definition | |
| 5.1.2 Missing data | |
| 5.1.3 Pooling of centers | |
| 5.2 Demographic and other background data | |
| 5.2.1 Basic description | |
| 5.3 IMP exposure, compliance | |
| 5.4 Medical history | |
| 5.5 Concomitant medication | |
| 5.6 Concomitant non-pharmacological measures, pre-medication | |
| 5.7 PK and Efficacy | |
| 5.7.2 Efficacy | |
| 5.7.3 Exploratory Endpoint | .19 |
| 5.8 Pharmacokinetics / Pharmacodynamics | .20 |
| 5.9 Surgeries | |
| 5.10 Safety | |
| 5.10.1 Adverse events | |
| 5.10.2 Vital signs | |
| 5.10.3 Safety laboratory variables | |
| 5.10.4 Other safety variables | |
| 5.11 Other variables | |
| 5.12 Interim analyses | |
| 6 Quality Control | |
| 7 References | |
| 8 Appendices | . 24 |



## STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.0 Date of Issue: 2017-04-26 

| 8.1 | Formulas for derived variables | 24 |
|---|---|---|
| 8.2 | Algorithm for the Overall Efficacy Assessment for Surgical Prophylaxis | 26 |
| | List of Tables, Listings, Figures | |




Date of Issue: 2017-04-26


### LIST OF ABBREVIATIONS

Abbreviation Description

ABR Annual Bleeding Rate

AE Adverse Event

ANOVA Analysis of Variance
AUC Area Under the Curve

AUC normalized for the administered dose

AUMC Area Under the Moment Curve

BE Bleeding Episode
BMI Body Mass Index

BW Body Weight

CD4 Cluster of Differentiation 4

CHR Chromogenic assay
CI Confidence Interval

CL Clearance

C<sub>max</sub> Maximum Plasma Concentration

CRF Case Report Form

CRO Contract Research Organization

CSR Clinical Study Report

DD Drug Dictionary (WHO Coding Thesaurus)

DBR Database Review

DMP Data Management Plan

DVP Data Validation Plan

ED Exposure Day

EDC Electronic Data Capture

EOT End of Trial

eCRF Electronic Case Report Form

FAS Full Analysis Set

FVIII Coagulation Factor VIII

FVIII:C Factor VIII-coagulant




Date of Issue: 2017-04-26


| Abbreviation | Desc | Description |
|--------------|------|-------------|

HJHS Hemophilia Joint Health Score

ICF Informed Consent Form

ID Identifier

IMP Investigational Medicinal Product

IRB Institutional Review Board

ITT Intention-To-Treat
IU International Unit

IV Intravenous

IVR Incremental in Vivo Recovery

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

MRT Mean Residence Time

N Number of Subjects/Observations

OS One-stage assay
PK Pharmacokinetic
POP Postoperative
PP Per-Protocol
PT Preferred Term

PTP Previously Treated Subject

QC Quality Control

SAE Serious Adverse Event

SAF Safety Analysis Set

SAP Statistical Analysis Plan

SAS Statistical Analysis Software package

SD Standard Deviation SOC System Organ Class

SOP Standard Operating Procedure

SABR Spontaneous Annualized Bleeding Rate

SURG Surgery analysis set




WHO

Date of Issue: 2017-04-26


| Abbreviation | Description |
|--------------|--------------------------------------------|
| $T_{1/2}$ | In Vivo Half-Life |
| TABR | Total Annualized Bleeding Rate |
| TEAE | Treatment Emergent Adverse Event |
| TLFs | Tables, Listings, Figures |
| $T_{max}$ | Time to Reach Maximum Plasma Concentration |
| TS | Trial Statistician |
| Vd | Volume of distribution |
| VWD | Von Willebrand Disease |
| VWF | Von Willebrand Factor |
| VWF:Ac | VWF activity |
| VWF:Ag | Von Willebrand Factor Antigen |

World Health Organization



|-----------------------------------------------|---------------|
| Version Number: 1.0 | Dags 10 of 27 |
| Date of Issue: 2017-04-26 | |

### 1 STUDY MATERIAL

The following material was considered for this SAP:

| Document | Version, Date |
|----------|-------------------------|
| Protocol | Version 1.0, 2017-04-26 |
| CRF | TBD |
| DMP | TBD |
| DVP | TBD |

### **2 STUDY INFORMATION**

### 2.1 Primary objective

The primary objective of this study is to determine the FVIII:C pharmacokinetics (PK) for *Wilate* in previously treated patients (PTP) with severe hemophilia A aged 1 to <12 years.

### 2.2 Secondary objective

The secondary objectives of this study are to:

- Determine the efficacy of *Wilate* in prophylactic treatment
- Determine the efficacy of *Wilate* in the treatment of breakthrough bleeding episodes (BEs)
- Calculate the FVIII:C incremental IVR of *Wilate* over time (at baseline, and at 3 and 6 months of treatment)
- Assess the association between AB0 blood type and the FVIII:C half-life of Wilate
- Assess the association between the VWF:Ag concentration and the FVIII:C half-life of *Wilate*
- Assess the safety and tolerability of Wilate
- Assess the immunogenicity of Wilate

### 2.3 Additional Objective:

An additional objective of this study is the descriptive efficacy of Wilate in surgical prophylaxis.




Date of Issue: 2017-04-26


### 2.4 Study design

This study is designed as a prospective, non-controlled, international, multi-center phase 3 study. Further details are given in the overview below:

### FLOW CHART FOR PK ASSESSMENT AND PROPHYLACTIC TREATMENT

| | Screen | PK<br>Visit | Pro<br>(starts wi | Follow-up<br>Contact<br>30 (±3) days<br>after | | | |
|---|---|---|---|---|---|---|---|
| | ing<br>Visit | | Day-14<br>Visit<br>(14–21<br>days) | Day-30<br>Visit<br>(±3<br>days) | 3-Month<br>Visit<br>(±2<br>weeks) | Study Completion (6-Month) Visit at 6 months (+2 weeks) | Study Com-<br>pletion<br>Visit |
| Informed consent | Х | | | | | | |
| Inclusion and exclusion criteria | Х | | | | | | |
| Demographics | Х | | | | | | |
| Weight | Х | x [1] | | | x [1] | x [1] | |
| Height | Х | | | | | | |
| Medical history (incl. FVIII treatment 6 months before screening) | x | | | | | | |
| Vital signs | Х | x [2] | | | x [4] | x [4] | |
| Physical examination | Х | | | | | х | |
| Routine safety laboratory | Х | x [3] | | | x [1] | x [4] | |
| Determination of CD4+ levels [8] | Х | | | | | | |
| Determination of AB0 blood group [9] | Х | | | | | | |
| HJHS, unless obtained within 3 months be-<br>fore screening | х | | | | | | |
| PK injection (50 ± 5 IU/kg) | | Х | | | | | |
| Blood sampling for FVIII:C (OS and CHR) for PK assessment | | x [5] | | | | | |
| IVR injection | | | | | Х | х | |
| Blood sampling for FVIII:C IVR (OS and CHR) | | | | | x [6] | x [6] | |
| Factor VIII inhibitor [10] | Х | x [1] | x [1] | x [1] | x [1] | x [1] | |
| VWF:Ag and VWF:Ac | | x [6] | x [1] | x [1] | x [6] | x [6] | |
| Parvovirus B19 antibodies | | x [1] | | | | x [7] | |
| Retention sample for possible virus marker testing | | x [1] | | | | | |
| Patient diary review | | | Х | Х | Х | х | |
| Adverse event monitoring | | Х | » | » | <b>»</b> | х | x [11] |
| Concomitant medications | Х | <b>»</b> | <b>»</b> | <b>»</b> | <b>»</b> | х | |

PK = pharmacokinetic, IVR = in vivo recovery, HJHS = Hemophilia Joint Health Score, OS = one-stage assay, CHR = chromogenic assay, VWF:Ag = von Willebrand factor antigen, VWF:Ac = VWF activity




Date of Issue: 2017-04-26


### LEGEND TO THE FLOW CHART FOR PK ASSESSMENT AND PROPHYLACTIC TREATMENT

- [1] Before injection
- [2] Before injection as well as 1 h (±5 min) and 48±2 h after injection
- [3] Before injection as well as 48±2 h after injection [local laboratory]
- [4] Before injection as well as 15±5 min after injection
- [5] Blood sampling within 1 h before injection and 15±5 min, 1 h (±5 min), 6 h (±30 min), 9±1 h, 24±2 h, 30±2 h, and 48±2 h after the end of injection [central laboratory]
- [6] Blood sampling within 1 h before injection as well as 15±5 min after the end of injection [central laboratory]
- [7] If first sample was negative for parvovirus B19 antibodies (sample to be taken before injection) [central laboratory]
- [8] CD4+ count to be repeated if interval between Screening Visit and first injection exceeds 30 days. To be included into the study, the patient's CD4+ count must be >200/μL (i.e., inclusion criterion no. 4).
- [9] Unless obtainable from patient's medical history
- [10] Blood sampling for inhibitor testing should preferably be done at the time of trough FVIII:C levels [central laboratory]
  In case of positive inhibitor results, inhibitor retesting using a second, separately drawn sample should be performed, preferably within 15 days of becoming aware of the positive result.
- [11] Documentation of any thromboembolic events only (to be documented on AE page)




Date of Issue: 2017-04-26


### FLOW CHART OF ASSESSMENTS FOR SURGICAL PROPHYLAXIS

| | Within | Within | Surg | ery | POP<br>day 1 | Any<br>POP<br>day | End of<br>POP<br>period | 3-8<br>weeks<br>after<br>surgery |
|---|---|---|---|---|---|---|---|---|
| | 12 hours<br>before<br>start | 3 hours<br>before<br>start | Intra-<br>opera-<br>tively | End<br>[1] | | | | |
| Body weight | Х | | | | | | | |
| Type of surgery | х | | | | | | | |
| Location of surgery | Х | | | | | | | |
| Severity of surgery | Х | | | | | | | |
| Expected duration of surgery | Х | | | | | | | |
| Expected average/ maximum blood loss during surgery | Х | | | | | | | |
| Actual duration of surgery | | | | х | | | | |
| Actual blood loss during surgery | | | | Х | | | | |
| Administration of IMP | | Х | (x) | (x) | (x) | (x) | (x) | |
| FVIII plasma levels | | # | (#) | (#) | # [2] | # | # | |
| VWF:Ag and VWF:Ac | | # | | | # [2] | # | # | |
| Presence of wound hematomas | | | | | х | Х | х | |
| Routine safety laboratory | Х | | | | (x) | (x) | (x) | |
| Vital signs | Х | | Х | | х | | | |
| Efficacy assessment | | | | S | | | Н | |
| Overall efficacy assessment | | | | | | | ı | |
| Factor VIII inhibitor [3] | | | | | | | | Х |
| Narrative of outcome | | | | | | | х | |
| Concomitant medications | throughout observation period | | | | | | | |
| Adverse event monitoring | throughout observation period | | | | | | | |

POP = postoperative, VWF:Ag = von Willebrand factor antigen, VWF:Ac = VWF activity

### 2.5 Planned sample size

Overall, 10 PTPs (5 patients aged 1 to <6 years of age and 5 patients aged 6 to <12 years) will be enrolled into this study. The aim is to obtain evaluable data on 8 patients who complete both the 2-day PK Phase and the 6-month Prophylactic Treatment Phase. Of the 8 evaluable patients, 4 patients must be 1 to <6 years of age, and another 4 patients must be 6 to <12 years of age. Enrolled patients will be replaced only if they do not complete the PK assessment.

The sample size of 10 pediatric patients to be enrolled was based on medical and regulatory reasoning. No statistical sample size estimation was performed.

<sup>()</sup> Optional

<sup>#</sup> Samples to be taken immediately before (≤ 30 min) and 30±15 min after IMP administration

<sup>[1]</sup> Time immediately after the last surgical suture

<sup>[2]</sup> For major surgeries, mandatory for the first 3 postoperative doses

<sup>[3]</sup> In case of positive inhibitor results, inhibitor retesting using a second, separately drawn sample should be performed, preferably within 15 days of becoming aware of the positive result.

S, performed by surgeon; H, performed by hematologist; I performed by Investigator



|-----------------------------------------------|---------------|
| Version Number: 1.0 | D 14 - 6 27 |
| Date of Issue: 2017-04-26 | |

### **3 GENERAL INFORMATION**

### 3.1 Background details

The data will be transferred to SAS from the Clinical Data Management System OPVERDI via a validated procedure. If applicable, external data will also be transferred to SAS for presentation of these data in the statistical analyses.

### 3.2 Deviations from the trial protocol with regard to statistical analyses

No deviations from the protocol are planned.

### 3.3 Individual protocol deviations

Any deviation from protocol will be discussed case by case before database lock whether the deviation has to be regarded as minor or as major (and therefore will lead to exclusion from particular analysis populations).

Examples for minor protocol violations may be deviations from scheduled investigation time.

Criteria for major protocol violations will at least include:

- Any substantial violation of in- or exclusion criteria.
- Use of concomitant medication that may interfere with the assessment of efficacy.

The final decision about the classification of individual protocol deviations and their consequences regarding assignment of subjects to analysis sets will be made during the data review meeting (DBR). A complete listing of protocol deviations and the judgment for assessment of subject disposition will be approved by the Sponsor and signed before database lock. All deviations along with the disposition of each subject will be recorded in a separate database member that will become part of the study database. A description of all major protocol violations will be included in the table part of the CSR.

### **4 ANALYSIS POPULATIONS**

The disposition of subjects will be displayed according to the following analysis populations:

- Safety (SAF) set
- Full Analysis set (FAS)
- Pharmacokinetic (PK) set
- Per-Protocol (PP) set
- Surgery (SURG) set



|-----------------------------------------------|---------------|
| Version Number: 1.0 | D 15 - 6 27 |
| Date of Issue: 2017-04-26 | |

### 4.1 Safety set

The safety (SAF) set will include all subjects who received at least one infusion of IMP.

### 4.2 Full analysis set

The **full analysis set (FAS)** defined according to the intention-to-treat (ITT) principle will include all enrolled subjects who received at least one infusion of IMP (after the initial PK visit).

### 4.3 Pharmacokinetic set

The **pharmacokinetic (PK) set** will include all patients for which a valid *Wilate* PK profile has been obtained.

### 4.4 Per-protocol set

The **per-protocol (PP) set**, i.e. a subset of the FAS, will exclude subjects with major protocol deviations which may have an impact on the evaluation of the primary study outcome parameter (major protocol deviations as defined during DBR).

### 4.5 Surgery set

The **surgery (SURG) set** will be a subset of the FAS, containing all subjects who underwent a surgical procedure treated with *Wilate* during their Prophylactic Treatment Phase.

### 4.6 Subgroup analyses

The analyses of the PK parameters and the efficacy endpoints 'efficacy of prophylactic treatment' and 'efficacy in treatment of breakthrough BEs' will be presented by age groups ('1 to <6 years' and '6 to <12 years').

### **5 STATISTICAL ANALYSES**

All statistical analyses will be performed using SAS® for Windows (Version 9.3 or later).

Descriptive statistics will always be given for the entire population.

The analysis of safety will be based on the SAF set.

Analysis of the PK properties of Wilate will be based on the PK set.

For secondary endpoints, FAS and PP analyses will be carried out, unless these analysis sets differ by no more than 1 patient from the FAS.

Analysis of the efficacy and safety of Wilate in surgeries will be based on the SURG set.

If not stated otherwise the following standard descriptive statistics will be presented:




Date of Issue: 2017-04-26


### Descriptive statistics for continuous data

Number of subjects (N), arithmetic mean, standard deviation (SD), minimum, lower quartile, median, upper quartile and maximum will be presented. Usually mean and quartiles will have 1 decimal more, SD 2 decimals more than the original values (as given with min, max); N has no decimals. These descriptive statistics will be determined for measured values and for differences to baseline.

### Descriptive statistics for categorical data

Absolute frequencies (N) will be presented with 0, relative frequencies (%) with 1 decimal. For changes from baseline, shift tables may be generated.

### Inferential statistics

If not stated otherwise all statistical tests will be performed as described in the corresponding sections below.

All p-values will be rounded to 4 decimals (p<0.0001 will be displayed, if the p-values are less than 0.0001). Statistical significance will be declared if the rounded p-value will be less than 0.05.

All confidence intervals (CI) will be derived two-sided and at a confidence probability of 1- $\alpha = 0.95$ .

### Listings

All subject data will be listed by subject. Identification variable will be the subject ID (composed of study, center and subject number separated by a hyphen, e.g. '30-01-01'. Any derived data listed will also be stored permanently and will be calculated as outlined in section 8.1 of this SAP.

### 5.1 Conventions

### 5.1.1 Baseline definition

Assessments at PK visit or at screening visit (in case the corresponding assessment is not scheduled at PK visit) are considered as baseline.

### 5.1.2 Missing data

In case of missing weight documentation data will be imputed using the Last Observation Carried Forward (LOCF) approach to calculate the dose per kg body weight (IU/kg). For calculation of PK parameters, missing measurements on a subject's PK profile will be handled according to the algorithms included in the PK software WinNonlin (version 7.0).

No further imputations for missing data will be performed.

Calculations pertaining to the derivation of annual bleeding rates will be based on documented time periods only.



|-----------------------------------------------|---------------|
| Version Number: 1.0 | Dags 17 of 27 |
| Date of Issue: 2017-04-26 | |

### 5.1.3 Pooling of centers

All tables will be presented in total over all participating countries and centers. The distribution of number of subjects per country and center will be presented in the disposition section of the report.

### 5.2 Demographic and other background data

### 5.2.1 Basic description

The disposition of subjects (cf. Section 4) will be tabulated for the entire population. Details on protocol deviations will be listed.

Discontinued subjects will be described by frequency distributions including the reasons and in individual listings.

Demographic data (age, weight, height, BMI, race, ethnic group) will be summarized in tables and presented for the SAF and FAS population. Other baseline or background data, e.g. disease-specific information, will comprise descriptive tables for the SAF and FAS population for the following variables:

- Blood group
- Last CD4+ level before enrolment
- VWF:Ag, VWF:Ac levels at PK visit
- FVIII inhibitor level
- Vital Signs (Systolic and diastolic blood pressure, pulse and body temperature) at screening
- Physical examination (normal/abnormal) at screening
- Hemophilia joint health score (HJHS) at screening
- Results of Parvovirus B19 antibodies at PK visit

The following background data will only be listed:

- Medical history (including FVIII treatment during the last 6 months before screening)
- Concomitant Medication

### 5.3 IMP exposure, compliance

Treatment will be administered prophylactically as defined in the protocol. Each home treatment will be recorded in the diary along with the reason for treatment (prophylaxis, bleeding, prevention of recurrent bleeding, prophylaxis after surgery or other reason). Treatments in context of IVR and PK measurements and surgeries will be documented in the patients notes. All treatments, from diary or patient's notes, will be transferred into the eCRF.

All IMP treatment details will be listed.



|-----------------------------------------------|---------------|
| Version Number: 1.0 | Dags 10 of 27 |
| Date of Issue: 2017-04-26 | |

### 5.4 Medical history

Data on medical history will be listed. Medical history will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Codes will be reviewed by a Medical Expert and approved by the sponsor before data base lock.

### 5.5 Concomitant medication

Any relevant medication taken at time of screening and all new medications taken by the subject during the study period are defined as 'Concomitant'. Any changes of medications during the study period will also be recorded.

All details of concomitant medications will be listed including, the route, dose, frequency, start and stop date and indication.

Medications will be coded using the WHO DD thesaurus in the version current at the time of database lock. Coding will be performed by the CRO and agreed upon with the sponsor before data base lock. (cf. DMP). For concomitant medications tables will show the frequencies of subjects by WHO DD preferred term.

### 5.6 Concomitant non-pharmacological measures, pre-medication

Not applicable.

### 5.7 PK and Efficacy

### 5.7.1 Pharmacokinetics

The primary objective of this study is the analysis of the PK profile of Wilate (refer to section 5.8).

### 5.7.2 Efficacy

All efficacy variables will be analyzed based on the FAS and additionally on the PP set, unless these analysis sets are identical.

Efficacy endpoints are:

- Efficacy of prophylactic treatment with *Wilate* based on the total annualized bleeding rate (TABR) as well as the spontaneous annualized bleeding rate (SABR)
- Efficacy of *Wilate* in the treatment of breakthrough BEs based on the proportion of BEs successfully treated with *Wilate* (successfully includes efficacy ratings assessed as either 'excellent' or 'good')
- Wilate consumption data (FVIII IU/kg per week and per month per subject) for prophylaxis




Date of Issue:

### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 

• Incremental IVR of *Wilate* over time (at baseline, and at 3 and 6 months of treatment) (refer to section 5.8)

### Efficacy of Prophylactic Treatment with Wilate

2017-04-26

The analysis of the efficacy of prophylactic treatment with *Wilate* will be statistically evaluated by presenting descriptive sampling statistics for the TABR and SABR, along with an exploratory 95% CI for the mean. TABR and SABR will be calculated as the total number of BEs or total number of spontaneous BEs, respectively, in the time period between first dose of IMP and the study completion visit, divided by the duration (in years) between first dose of IMP and the study completion visit. Surgery periods, and BEs occurring within these periods, will be excluded from the calculation of annual bleeding rates

### Efficacy in the Treatment of Breakthrough BEs

To assess the hemostatic efficacy of *Wilate* in the treatment of breakthrough bleedings, a frequency distribution of all such BEs being successfully treated will be presented, along with an exploratory 95% CI.

Primarily, all obtained data on treatment characteristics (IMP dosages, frequencies, total consumption) and BEs (duration, frequency, efficacy assessment) will be described by providing summary statistics.

In general, the efficacy of bleeding episodes will also be presented by type (spontaneous, traumatic, postoperative, other), sites (nose, oral cavity, knee, ankle, elbow, arm, leg, intestinal and other. In addition, knee, ankle and elbow sites will be summarized as site 'joint') and severity (minor, moderate, major, life-threatening).

### Analysis of Other Secondary Endpoints

The statistical analysis of other secondary endpoints will be descriptive, including exploratory 95% CIs for the location parameters.

### 5.7.3 Exploratory Endpoint

An exploratory endpoint of this study is the descriptive efficacy of *Wilate* in surgical prophylaxis (for details see section 5.9).



|-----------------------------------------------|---------------|
| Version Number: 1.0 | Dags 20 of 27 |
| Date of Issue: 2017-04-26 | |

### 5.8 Pharmacokinetics / Pharmacodynamics

For Pharmacokinetics and IVR assessments FVIII:C will be measured by both, the chromogenic (CHR) and one-stage assay (OS) and analyzed based on actual IMP potency (refer to section 8.1).

The PK profiles of *Wilate* and the PK parameters derived from them will be summarized by descriptive statistics as well as the presentation of concentration vs. time plots based on the PK set. In the analysis of the PK profiles geometric means and standard deviations will be presented in addition to the arithmetic means and standard deviations.

The following PK parameter will be derived and presented using a non-compartment model:

- Area under the curve (AUC) and AUC normalized for the administered dose (AUC<sub>norm</sub>)
- FVIII in vivo half-life  $(T_{1/2})$
- Maximum plasma concentration (C<sub>max</sub>)
- Time to reach maximum plasma concentration (T<sub>max</sub>)
- Mean residence time (MRT)
- Volume of distribution (Vd)
- Clearance (CL)
- Incremental in vivo recovery (IVR)

Analysis of variance (ANOVA) will be used in an exploratory sense to assess a possible association between AB0 blood type, VWF:Ag, and the FVIII:C half-life of *Wilate*.

Incremental IVR will be calculated from FVIII:C plasma levels measured before injection and peak levels obtained in the 15-min post-injection sample using actual IMP potencies. The results of the IVR assessments over time will be analyzed in summary tables for each time point and their differences to baseline along with 95% CIs for the mean differences.

### 5.9 Surgeries

Efficacy in surgical prophylaxis will be analyzed descriptively, presenting summary tables and listing on all aspects of surgical treatment and procedures as well as efficacy ratings.

The following surgery-related parameters will be presented:

- Number of minor and major surgeries
- Location, severity (minor or major, for definitions see protocol), and type (planned or emergency) of surgery
- Expected and actual duration of surgical procedure
- Expected and actual blood loss
- Pre-, intra-, and/or postoperative IMP administration data (only listed)



### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.0 Date of Issue: 2017-04-26 

- Pre-, intra-, and postoperative FVIII plasma levels (only listed)
- VWF:Ag and VWF:Ac (descriptive statistics including changes to pre-infusion)
- Frequency and amount of blood transfusion requirements
- Presence of wound hematomas and whether or not they require surgical evacuation (only listed)
- Assessment of efficacy of surgical prophylaxis:
  - 1. at the end of surgery by the surgeon
  - 2. at end of the postoperative period by the hematologist
  - 3. Overall efficacy taking both the intra- and postoperative assessments into account assessed by the Investigator.
- Number of successively treated surgeries ('excellent' or 'good' overall efficacy rating)
- Concomitantly administered products (only listed)
- Narrative describing the outcome and efficacy of the intervention (only listed)
- Inhibitor testing (within 3–8 weeks after the end of the surgery, this visit may coincide with another study visit with scheduled inhibitor testing)

### 5.10 Safety

All safety analyses will be based on the SAF population.

The analysis of safety will include the occurrence of AEs, the results of the safety laboratory tests, immunogenicity measurements and the occurrence of parvovirus B19 seroconversions.

### 5.10.1 Adverse events

Adverse events (AEs) will be coded by the CRO according to the latest Medical Dictionary for Regulatory Activities (MedDRA). Coding will be agreed upon with the Sponsor before database lock (cf. DMP).

All adverse events recorded since signing of the informed consent form (ICF) will be listed in appendix 16.2 of the report differentiating by treatment emergent and non-treatment emergent events. This includes also post-study serious adverse events (SAEs) which occurred up to 4 weeks after the last IMP administration (not monitored proactively), thromboembolic events monitored proactively by performing a Follow-up Contact 30 days after the completion visit as well as safety relevant information on drug overdosing, drug interactions and medication errors.

The analysis will include only treatment-emergent adverse events (TEAEs), i.e. all documented AEs that started or worsened after the start of IMP infusion. It is assumed that for each increase in intensity of an AE a new entry of the AE will be done by the investigator; hence such cases will be analyzed like different phases of the same AE.



## STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.0 Date of Issue: 2017-04-26 

A descriptive analysis will be performed. Incidences will be presented by primary system organ classes (SOC) and incidences of PT within primary SOC sorted according to the Internationally Agreed Order.

Multiple counts within a PT or SOC (repeated or different included terms or changes in descriptors) will be counted only once for the calculation of incidences.

Global incidences will be calculated for:

- All TEAE irrespective of the causality assessment
- Related TEAEs ('Probably' or 'Possible')
- TEAEs by worst severity
- Serious TEAEs

A listing of "special cases" containing subject identification, age, sex, AE descriptors, start and end of treatment will be prepared for the following types of TEAEs:

- Serious adverse events (SAE)
- Adverse events which led to death
- Adverse events which led to discontinuation

Serious non-treatment emergent AEs will be listed separately.

### 5.10.2 Vital signs

Vital signs parameters (systolic/diastolic blood pressure, pulse, body weight, respiratory rates, body temperature) will be assessed at screening, PK visit, after 3 months at study completion visits and during surgery.

Descriptive analyses of values will be performed and changes from baseline will be analyzed for vital signs parameters at visits.

### 5.10.3 Safety laboratory variables

The analysis of the safety parameters (lab values for Hematology and Clinical chemistry) recorded during visits (screening, PK visit, 3-month and study completion visits) and at surgery will be purely descriptive and presented as summary tables or listings.

Time profiles of the safety laboratory parameters will be analyzed by presenting sampling statistics for the values as well as their difference to baseline at each time point. Additionally, frequency tables for values outside the normal ranges will be presented.

Similarly, time profiles of FVIII inhibitor testing results will be analyzed by presenting sampling statistics for the values as well as frequency tables for positive findings, along with 95% Pearson-Clopper CIs.




The thromboembolic risk will be monitored by determination of VWF:Ag and VWF:Ac during the study and especially postoperatively. Descriptive statistics including changes to preinfusion will be presented by visit and timepoint (with 95% CI) for visits or by operative day and timepoint for surgeries, respectively.

To assess the viral safety of *Wilate* incidences of parvovirus B19 seroconversions between baseline and end of study will be estimated along with 95% Pearson-Clopper CIs.

### 5.10.4 Other safety variables

Other safety parameters (e.g., changes in physical examination findings) will be analyzed by summary tables or listings. All abnormal findings from the physical examination will be listed.

The analysis of the safety parameters recorded during surgery (lab values) will be purely descriptive and presented as summary tables or listings.

### 5.11 Other variables

Not applicable.

### 5.12 Interim analyses

Not applicable.

### **6 QUALITY CONTROL**

The responsible project manager will review the SAP before it is provided to the Sponsor for review. The SAP will be signed off only when approval from the Sponsor's representative is received.

Log files of all SAS® programs needed for analysis will be checked for errors, warnings and suspicious notes by the statistical programmer. All findings will be either eliminated or commented upon. The final version of each program will be stored along with its log file in the electronic archive.

All programs will be validated by the author.

The agreement of the program outputs with the SAP, their consistency and plausibility will be checked by the TS. Moreover, the TS will review the outputs regarding completeness, readability and comprehensibility.

### **7 REFERENCES**

No specific references were used.



|-----------------------------------------------|------------|---------------|
| Version Number: | 1.0 | D 24 - 627 |
| Date of Issue: | 2017-04-26 | |

### 8 APPENDICES

### 8.1 Formulas for derived variables

| Variable | Description |
|---|---|
| Actual potency | Potency of IMP (IU) based on central laboratory measurements of FVIII content by two assay methods: CHR (chromogenic) and OS (one-stage). The analysis of PK and IVR assessment will be based on actual potencies |
| Durations be- | Later date minus earlier date plus 1, expressed in days. (Remark: Du- |
| Annual bleeding rate | ration will be 1, if both dates are the same.) Number of bleeding / (last date of IMP – first date of IMP + 1)/365.25 |
| AUC | Area under the curve from baseline to infinity |
| | $AUC = \sum \left( \frac{(C_n + C_{n+1})}{2} \cdot \Delta t \right) + \frac{C_{last}}{K}$ |
| | (C <sub>last</sub> is the last available measurement) |
| AUC <sub>norm</sub> | AUC normalized for the administered dose |
| AUMC | Area under the moment curve (from baseline to infinity) |
| | $AUMC = \sum \left( \frac{(t_n \cdot C_n + t_{n+1}C_{n+1})}{2} \cdot \Delta t \right) + \frac{C_{last}}{K^2} + \frac{t_{last} \cdot C_{last}}{K}$ |
| CL | Clearance |
| | $CL = \frac{D}{AUC}$ |
| | where $D$ is the actual dose administered (see remark above) |
| $C_0$ | FVIII concentration before IPM administration |
| C <sub>max</sub> | Maximal measured concentration after end of IMP infusion (peak concentration) |
| ED | Exposure day = each calendar day the subject received IMP |
| Incremental re-<br>covery (IVR) | $IVR = \frac{(C_{\text{max}} - C_0) \cdot BW}{D}$ |
| | where BW stands for the body weight in kg and D is the dose according to the actual potency of the FVIII concentrate as described in above |
| Labelled potency | Potency of IMP (IU) based on label of vial (IU). |




Date of Issue: 2017-04-26


| | Dosing analyses will be based on labelled potency |
|---|---|
| MRT | Mean residence time |
| | $MRT = \frac{AUMC}{AUC}$ |
| Success (for | Excellent or good efficacy rating |
| bleeding epi- | |
| sodes and sur- | |
| geries) | |
| $T_{1/2}$ | In vivo half-life |
| | using linear regression on the terminal phase of the logarithm of the concentration; |
| | $T_{\frac{1}{2}} = \frac{\ln(2)}{K}$ |
| | (where <i>K</i> , the elimination rate constant, is determined as the slope of the regression line) |
| T <sub>max</sub> | Time to reach maximum plasma concentration (Timing starts at end of infusion) |
| Vd | Volume of distribution |
| | $Vd = CL \cdot MRT$ |




Date of Issue: 2017-04-26


### 8.2 Algorithm for the Overall Efficacy Assessment for Surgical Prophylaxis

The evaluation of overall efficacy of the treatment in surgeries based on the intraoperative and postoperative assessment is defined as described below:

| Intraoperative | Postoperative assessment | | | |
|----------------|--------------------------|----------|----------|----------|
| assessment | Excellent | Good | Moderate | None |
| Excellent | Excellent | Good | Good | Moderate |
| Good | Good | Good | Moderate | Moderate |
| Moderate | Good | Moderate | Moderate | None |
| None | Good | Moderate | None | None |



### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30


Date of Issue: 2017-04-26


### 8.3 List of Tables, Listings, Figures

A complete lists of tables, listings figures (TLFs) will be given in a separate document which can be updated without updating the SAP. The list will serve as a reference for both the Sponsor, the trial statistician and the statistical programmer and includes the totality of statistical output to be produced. Therefore, this list will be approved by both parties before commencing the statistical programming.

All output will be headed with an appropriate heading specifying the study ID and abbreviated study title.

All output will be dated and have page numbers in the form 'Page [x / y]' where x denotes the current page within an output and y the total number of pages of that output.

All statistical output will identify the underlying analysis populations and indicate the number of subjects / events in this population (N) and the number of subject/events actually contributing to the particular output (n). All statistical output will be presented per treatment group and in total (if applicable).

All subject listings will contain additionally to the subject identification the analysis population and the treatment group.




Version Number: 1.1

Date of Issue: 2017-05-24


| Sponsor: | Octapharma AG |
|---|---|
| Title of Protocol: | Clinical Study to Investigate the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of <i>Wilate</i> in Previously Treated Pediatric Patients with Severe Hemophilia A |
| Protocol Version/Date: | Version 1.0 / 2017-05-15 |
| CRF Version: | TBD |
| Supersedes SAP Version: | None |


This document contains confidential information which must not be disclosed to anyone other than the involved CRO. This information should not be used for any purpose other than the evaluation of the clinical investigation without prior written consent of Octapharma.

No part of this document may be reproduced or stored in a retrieval system or transmitted in any other form or by any other means.



### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30


Date of Issue: 2017-05-24


### **Document authorization**





|-----------------------------------------------|------------|--------------|
| Version Number: 1.1 | | D 2 627 |
| Date of Issue: | 2017-05-24 | |

### Consistency check with the Protocol (one option to be selected)

This is to confitm that as part of the SAP finalization consistency check with the current protocol / protocol amendment was performed by the trial statistician, and no changes to the protocol (statistical section) are required

- D Changes to the analysis principles were required, and the responsible team has confirmed commitment to update the study protocol
- D Changes to the analysis principles were required (as outlined in revision history section of this SAP), however it was not feasible to update the study protocol, for the reason





|-----------------------------------------------|--------------|
| Version Number: 1.1 | D 4 - 6 27 |
| Date of Issue: 2017-05-24 | |

### Change control

| Date | Author | Reason | Version |
|---|---|---|---|
| 2017-04-26 | | | 1.0 |
| 2017-05-24 | | SAP adapted to protocol version 01, 15-May-2017 | 1.1 |




Date of Issue: 2017-05-24


### TABLE OF CONTENTS

| Document authorization | |
|---|---|
| Consistency check with the Protocol (one option to be selected) | |
| Change control | |
| Table of contents | |
| List of abbreviations | |
| 1 Study material | |
| 2 Study information | |
| 2.1 Primary objective | |
| 2.2 Secondary objective | |
| 2.3 Additional Objective: | |
| 2.4 Study design | |
| 2.5 Planned sample size | |
| 3 General Information | |
| 3.1 Background details | 14 |
| 3.2 Deviations from the trial protocol with regard to statistical analyses | .14 |
| 3.3 Individual protocol deviations | 14 |
| 4 Analysis Populations | . 14 |
| 4.1 Safety set | 15 |
| 4.2 Full analysis set | .15 |
| 4.3 Pharmacokinetic set | |
| 4.4 Per-protocol set | |
| 4.5 Surgery set | |
| 4.6 Subgroup analyses | |
| 5 Statistical Analyses | |
| 5.1 Conventions | |
| 5.1.1 Baseline definition. | |
| 5.1.2 Missing data | |
| 5.1.3 Pooling of centers | |
| 5.2 Demographic and other background data | |
| 5.2.1 Basic description | |
| 5.3 IMP exposure, compliance | |
| 5.4 Medical history | |
| 5.5 Concomitant medication | |
| 5.6 Concomitant non-pharmacological measures, pre-medication | |
| 5.7 PK and Efficacy | |
| 5.7.2 Efficacy | |
| 5.7.2 Efficacy | |
| 5.8 Pharmacokinetics / Pharmacodynamics | |
| 5.9 Surgeries | |
| 5.10 Safety | |
| 5.10.1 Adverse events | |
| 5.10.2 Vital signs | |
| 5.10.3 Safety laboratory variables | |
| 5.10.4 Other safety variables | |
| 5.11 Other variables | |
| 5.12 Interim analyses | |
| 6 Quality Control | |
| 7 References | |
| 8 Appendices | |



# STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.1 Date of Issue: 2017-05-24 

| 8.1 | Formulas for derived variables | 24 |
|---|---|---|
| 8.2 | Algorithm for the Overall Efficacy Assessment for Surgical Prophylaxis | 26 |
| | List of Tables, Listings, Figures | |




Date of Issue: 2017-05-24


### LIST OF ABBREVIATIONS

Abbreviation Description

ABR Annual Bleeding Rate

AE Adverse Event

ANOVA Analysis of Variance
AUC Area Under the Curve

AUC normalized for the administered dose

AUMC Area Under the Moment Curve

BE Bleeding Episode
BMI Body Mass Index

BW Body Weight

CD4 Cluster of Differentiation 4

CHR Chromogenic assay
CI Confidence Interval

CL Clearance

C<sub>max</sub> Maximum Plasma Concentration

CRF Case Report Form

CRO Contract Research Organization

CSR Clinical Study Report

DD Drug Dictionary (WHO Coding Thesaurus)

DBR Database Review

DMP Data Management Plan

DVP Data Validation Plan

ED Exposure Day

EDC Electronic Data Capture

EOT End of Trial

eCRF Electronic Case Report Form

FAS Full Analysis Set

FVIII Coagulation Factor VIII

FVIII:C Factor VIII-coagulant




Date of Issue: 2017-05-24 

| Abbreviation | Description | |
|--------------|-------------|---------|
| LILLIC | т т | 1 '1' т |

Hemophilia Joint Health Score HJHS

**ICF** Informed Consent Form

ID Identifier

**IMP** Investigational Medicinal Product

Institutional Review Board **IRB** 

Intention-To-Treat TTT IU International Unit

IV Intravenous

IVR Incremental in Vivo Recovery

Last Observation Carried Forward **LOCF** 

MedDRA Medical Dictionary for Regulatory Activities

MRT Mean Residence Time

Number of Subjects/Observations Ν

Preferred Term

OS One-stage assay PΚ Pharmacokinetic POP Postoperative PР Per-Protocol РΤ

PTP Previously Treated Subject

QC Quality Control

SAE Serious Adverse Event

SAF Safety Analysis Set

SAP Statistical Analysis Plan

SAS Statistical Analysis Software package

Standard Deviation SD System Organ Class SOC

SOP Standard Operating Procedure

**SABR** Spontaneous Annualized Bleeding Rate

**SURG** Surgery analysis set



Date of Issue: 2017-05-24


| Abbreviation | Description |
|--------------|--------------------------------------------|
| $T_{1/2}$ | In Vivo Half-Life |
| TABR | Total Annualized Bleeding Rate |
| TEAE | Treatment Emergent Adverse Event |
| TLFs | Tables, Listings, Figures |
| $T_{max}$ | Time to Reach Maximum Plasma Concentration |
| TS | Trial Statistician |
| Vd | Volume of distribution |
| VWD | Von Willebrand Disease |
| VWF | Von Willebrand Factor |
| VWF:Ac | VWF activity |
| VWF:Ag | Von Willebrand Factor Antigen |
| WHO | World Health Organization |



|-----------------------------------------------|---------------|
| Version Number: 1.1 | Dags 10 of 27 |
| Date of Issue: 2017-05-24 | |

### 1 STUDY MATERIAL

The following material was considered for this SAP:

| Document | Version, Date |
|----------|-------------------------|
| Protocol | Version 1.0, 2017-04-26 |
| CRF | TBD |
| DMP | TBD |
| DVP | TBD |

### **2 STUDY INFORMATION**

### 2.1 Primary objective

The primary objective of this study is to determine the FVIII:C pharmacokinetics (PK) for *Wilate* in previously treated patients (PTP) with severe hemophilia A aged 1 to <12 years.

### 2.2 Secondary objective

The secondary objectives of this study are to:

- Determine the efficacy of *Wilate* in prophylactic treatment
- Determine the efficacy of *Wilate* in the treatment of breakthrough bleeding episodes (BEs)
- Calculate the FVIII:C incremental IVR of Wilate over time (at baseline, and at 3 and 6 months of treatment)
- Assess the association between AB0 blood type and the FVIII:C half-life of Wilate
- Assess the association between the VWF:Ag concentration and the FVIII:C half-life of Wilate
- Assess the safety and tolerability of Wilate
- Assess the immunogenicity of Wilate

### 2.3 Additional Objective:

An additional objective of this study is the descriptive efficacy of Wilate in surgical prophylaxis.




Date of Issue: 2017-05-24


### 2.4 Study design

This study is designed as a prospective, non-controlled, international, multi-center phase 3 study. Further details are given in the overview below:

### FLOW CHART FOR PK ASSESSMENT AND PROPHYLACTIC TREATMENT

| | Screen | PK<br>Visit | Prophylactic Treatment Phase (starts with first prophylactic injection of <i>Wilate</i> after the PK Visit) | | | | Follow-up<br>Contact<br>30 (±3) days<br>after |
|---|---|---|---|---|---|---|---|
| | ing<br>Visit | | Day-14<br>Visit<br>(14–21<br>days) | Day-30<br>Visit<br>(±3<br>days) | 3-Month<br>Visit<br>(±2<br>weeks) | Study Completion (6-Month) Visit at 6 months (+2 weeks) | Study Com-<br>pletion<br>Visit |
| Informed consent | Х | | | | | | |
| Inclusion and exclusion criteria | Х | | | | | | |
| Demographics | Х | | | | | | |
| Weight | Х | x [1] | | | x [1] | x [1] | |
| Height | Х | | | | | | |
| Medical history (incl. FVIII treatment 6 months before screening) | x | | | | | | |
| Vital signs | Х | x [2] | | | x [4] | x [4] | |
| Physical examination | Х | | | | | х | |
| Routine safety laboratory | Х | x [3] | | | x [1] | x [4] | |
| Determination of CD4+ levels [8] | Х | | | | | | |
| Determination of AB0 blood group [9] | Х | | | | | | |
| HJHS, unless obtained within 3 months be-<br>fore screening | х | | | | | | |
| PK injection (50 ± 5 IU/kg) | | Х | | | | | |
| Blood sampling for FVIII:C (OS and CHR) for PK assessment | | x [5] | | | | | |
| IVR injection | | | | | Х | х | |
| Blood sampling for FVIII:C IVR (OS and CHR) | | | | | x [6] | x [6] | |
| Factor VIII inhibitor [10] | Х | x [1] | x [1] | x [1] | x [1] | x [1] | |
| VWF:Ag and VWF:Ac | | x [6] | x [1] | x [1] | x [6] | x [6] | |
| Parvovirus B19 antibodies | | x [1] | | | | x [7] | |
| Retention sample for possible virus marker testing | | x [1] | | | | | |
| Patient diary review | | | Х | Х | Х | х | |
| Adverse event monitoring | | Х | » | » | <b>»</b> | х | x [11] |
| Concomitant medications | Х | <b>»</b> | <b>»</b> | <b>»</b> | <b>»</b> | х | |

PK = pharmacokinetic, IVR = in vivo recovery, HJHS = Hemophilia Joint Health Score, OS = one-stage assay, CHR = chromogenic assay, VWF:Ag = von Willebrand factor antigen, VWF:Ac = VWF activity




Date of Issue: 2017-05-24


### LEGEND TO THE FLOW CHART FOR PK ASSESSMENT AND PROPHYLACTIC TREATMENT

- [1] Before injection
- [2] Before injection as well as 1 h (±5 min) and 48±2 h after injection
- [3] Before injection as well as 48±2 h after injection [local laboratory]
- [4] Before injection as well as 15±5 min after injection
- [5] Blood sampling within 1 h before injection and 15±5 min, 1 h (±5 min), 6 h (±30 min), 9±1 h, 24±2 h, and 48±2 h after the end of injection [central laboratory]
- [6] Blood sampling within 1 h before injection as well as 15±5 min after the end of injection [central laboratory]
- [7] If first sample was negative for parvovirus B19 antibodies (sample to be taken before injection) [central laboratory]
- [8] CD4+ count to be repeated if interval between Screening Visit and first injection exceeds 30 days. To be included into the study, the patient's CD4+ count must be >200/μL (i.e., inclusion criterion no. 4).
- [9] Unless obtainable from patient's medical history
- [10] Blood sampling for inhibitor testing should preferably be done at the time of trough FVIII:C levels [central laboratory]
  In case of positive inhibitor results, inhibitor retesting using a second, separately drawn sample should be performed, preferably within 15 days of becoming aware of the positive result.
- [11] Documentation of any thromboembolic events only (to be documented on AE page)




Date of Issue: 2017-05-24


### FLOW CHART OF ASSESSMENTS FOR SURGICAL PROPHYLAXIS

| | Within | Within | Surg | ery | | | End of<br>POP<br>period | 3-8<br>weeks<br>after<br>surgery |
|---|---|---|---|---|---|---|---|---|
| | 12 hours<br>before<br>start | 3 hours<br>before<br>start | Intra-<br>opera-<br>tively | End<br>[1] | POP<br>day 1 | Any<br>POP<br>day | | |
| Body weight | х | | | | | | | |
| Type of surgery | Х | | | | | | | |
| Location of surgery | Х | | | | | | | |
| Severity of surgery | Х | | | | | | | |
| Expected duration of surgery | Х | | | | | | | |
| Expected average/ maximum blood loss during surgery | Х | | | | | | | |
| Actual duration of surgery | | | | х | | | | |
| Actual blood loss during surgery | | | | х | | | | |
| Administration of IMP | | Х | (x) | (x) | (x) | (x) | (x) | |
| FVIII plasma levels | | # | (#) | (#) | # [2] | # | # | |
| VWF:Ag and VWF:Ac | | # | | | # [2] | # | # | |
| Presence of wound hematomas | | | | | х | Х | х | |
| Routine safety laboratory | Х | | | | (x) | (x) | (x) | |
| Vital signs | Х | | Х | | х | | | |
| Efficacy assessment | | | | S | | | Н | |
| Overall efficacy assessment | | | | | | | | |
| Factor VIII inhibitor [3] | | | | | | | | Х |
| Narrative of outcome | x | | | | | | | |
| Concomitant medications | throughout observation period | | | | | | | |
| Adverse event monitoring | throughout observation period | | | | | | | |

POP = postoperative, VWF:Ag = von Willebrand factor antigen, VWF:Ac = VWF activity

### 2.5 Planned sample size

Overall, 10 PTPs (5 patients aged 1 to <6 years of age and 5 patients aged 6 to <12 years) will be enrolled into this study. The aim is to obtain evaluable data on 8 patients who complete both the 2-day PK Phase and the 6-month Prophylactic Treatment Phase. Of the 8 evaluable patients, 4 patients must be 1 to <6 years of age, and another 4 patients must be 6 to <12 years of age. Enrolled patients will be replaced only if they do not complete the PK assessment.

The sample size of 10 pediatric patients to be enrolled was based on medical and regulatory reasoning. No statistical sample size estimation was performed.

<sup>()</sup> Optional

<sup>#</sup> Samples to be taken immediately before (≤ 30 min) and 30±15 min after IMP administration

<sup>[1]</sup> Time immediately after the last surgical suture

<sup>[2]</sup> For major surgeries, mandatory for the first 3 postoperative doses

<sup>[3]</sup> In case of positive inhibitor results, inhibitor retesting using a second, separately drawn sample should be performed, preferably within 15 days of becoming aware of the positive result.

S, performed by surgeon; H, performed by hematologist; I performed by Investigator



### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.1 Date of Issue: 2017-05-24 

### **3 GENERAL INFORMATION**

### 3.1 Background details

The data will be transferred to SAS from the Clinical Data Management System OPVERDI via a validated procedure. If applicable, external data will also be transferred to SAS for presentation of these data in the statistical analyses.

### 3.2 Deviations from the trial protocol with regard to statistical analyses

No deviations from the protocol are planned.

### 3.3 Individual protocol deviations

Any deviation from protocol will be discussed case by case before database lock whether the deviation has to be regarded as minor or as major (and therefore will lead to exclusion from particular analysis populations).

Examples for minor protocol violations may be deviations from scheduled investigation time.

Criteria for major protocol violations will at least include:

- Any substantial violation of in- or exclusion criteria.
- Use of concomitant medication that may interfere with the assessment of efficacy.

The final decision about the classification of individual protocol deviations and their consequences regarding assignment of subjects to analysis sets will be made during the data review meeting (DBR). A complete listing of protocol deviations and the judgment for assessment of subject disposition will be approved by the Sponsor and signed before database lock. All deviations along with the disposition of each subject will be recorded in a separate database member that will become part of the study database. A description of all major protocol violations will be included in the table part of the CSR.

### **4 ANALYSIS POPULATIONS**

The disposition of subjects will be displayed according to the following analysis populations:

- Safety (SAF) set
- Full Analysis set (FAS)
- Pharmacokinetic (PK) set
- Per-Protocol (PP) set
- Surgery (SURG) set




### 4.1 Safety set

The safety (SAF) set will include all subjects who received at least one infusion of IMP.

### 4.2 Full analysis set

The **full analysis set (FAS)** defined according to the intention-to-treat (ITT) principle will include all enrolled subjects who received at least one infusion of IMP (after the initial PK visit).

### 4.3 Pharmacokinetic set

The **pharmacokinetic (PK)** set will include all patients for which a valid *Wilate* PK profile has been obtained.

### 4.4 Per-protocol set

The per-protocol (PP) set, i.e. a subset of the FAS, will exclude subjects with major protocol deviations which may have an impact on the evaluation of the primary study outcome parameter (major protocol deviations as defined during DBR).

### 4.5 Surgery set

The **surgery (SURG) set** will be a subset of the FAS, containing all subjects who underwent a surgical procedure treated with *Wilate* during their Prophylactic Treatment Phase.

### 4.6 Subgroup analyses

The analyses of the PK parameters and the efficacy endpoints 'efficacy of prophylactic treatment' and 'efficacy in treatment of breakthrough BEs' will be presented by age groups ('1 to <6 years' and '6 to <12 years').

### **5 STATISTICAL ANALYSES**

All statistical analyses will be performed using SAS® for Windows (Version 9.3 or later).

Descriptive statistics will always be given for the entire population.

The analysis of safety will be based on the SAF set.

Analysis of the PK properties of Wilate will be based on the PK set.

For secondary endpoints, FAS and PP analyses will be carried out, unless these analysis sets differ by no more than 1 patient from the FAS.

Analysis of the efficacy and safety of Wilate in surgeries will be based on the SURG set.

If not stated otherwise the following standard descriptive statistics will be presented:




Date of Issue: 2017-05-24


### Descriptive statistics for continuous data

Number of subjects (N), arithmetic mean, standard deviation (SD), minimum, lower quartile, median, upper quartile and maximum will be presented. Usually mean and quartiles will have 1 decimal more, SD 2 decimals more than the original values (as given with min, max); N has no decimals. These descriptive statistics will be determined for measured values and for differences to baseline.

### Descriptive statistics for categorical data

Absolute frequencies (N) will be presented with 0, relative frequencies (%) with 1 decimal. For changes from baseline, shift tables may be generated.

### Inferential statistics

If not stated otherwise all statistical tests will be performed as described in the corresponding sections below.

All p-values will be rounded to 4 decimals (p<0.0001 will be displayed, if the p-values are less than 0.0001). Statistical significance will be declared if the rounded p-value will be less than 0.05.

All confidence intervals (CI) will be derived two-sided and at a confidence probability of 1- $\alpha = 0.95$ .

### Listings

All subject data will be listed by subject. Identification variable will be the subject ID (composed of study, center and subject number separated by a hyphen, e.g. '30-01-01'. Any derived data listed will also be stored permanently and will be calculated as outlined in section 8.1 of this SAP.

### 5.1 Conventions

### 5.1.1 Baseline definition

Assessments at PK visit or at screening visit (in case the corresponding assessment is not scheduled at PK visit) are considered as baseline.

### 5.1.2 Missing data

In case of missing weight documentation data will be imputed using the Last Observation Carried Forward (LOCF) approach to calculate the dose per kg body weight (IU/kg). For calculation of PK parameters, missing measurements on a subject's PK profile will be handled according to the algorithms included in the PK software WinNonlin (version 7.0).

No further imputations for missing data will be performed.

Calculations pertaining to the derivation of annual bleeding rates will be based on documented time periods only.



|-----------------------------------------------|
| Date of Issue: 2017-05-24 |

### 5.1.3 Pooling of centers

All tables will be presented in total over all participating countries and centers. The distribution of number of subjects per country and center will be presented in the disposition section of the report.

### 5.2 Demographic and other background data

### 5.2.1 Basic description

The disposition of subjects (cf. Section 4) will be tabulated for the entire population. Details on protocol deviations will be listed.

Discontinued subjects will be described by frequency distributions including the reasons and in individual listings.

Demographic data (age, weight, height, BMI, race, ethnic group) will be summarized in tables and presented for the SAF and FAS population. Other baseline or background data, e.g. disease-specific information, will comprise descriptive tables for the SAF and FAS population for the following variables:

- Blood group
- Last CD4+ level before enrolment
- VWF:Ag, VWF:Ac levels at PK visit
- FVIII inhibitor level
- Vital Signs (Systolic and diastolic blood pressure, pulse and body temperature) at screening
- Physical examination (normal/abnormal) at screening
- Hemophilia joint health score (HJHS) at screening
- Results of Parvovirus B19 antibodies at PK visit

The following background data will only be listed:

- Medical history (including FVIII treatment during the last 6 months before screening)
- Concomitant Medication

### 5.3 IMP exposure, compliance

Treatment will be administered prophylactically as defined in the protocol. Each home treatment will be recorded in the diary along with the reason for treatment (prophylaxis, bleeding, prevention of recurrent bleeding, prophylaxis after surgery or other reason). Treatments in context of IVR and PK measurements and surgeries will be documented in the patients notes. All treatments, from diary or patient's notes, will be transferred into the eCRF.

All IMP treatment details will be listed.



|-----------------------------------------------|
| Date of Issue: 2017-05-24 |

### 5.4 Medical history

Data on medical history will be listed. Medical history will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Codes will be reviewed by a Medical Expert and approved by the sponsor before data base lock.

### 5.5 Concomitant medication

Any relevant medication taken at time of screening and all new medications taken by the subject during the study period are defined as 'Concomitant'. Any changes of medications during the study period will also be recorded.

All details of concomitant medications will be listed including, the route, dose, frequency, start and stop date and indication.

Medications will be coded using the WHO DD thesaurus in the version current at the time of database lock. Coding will be performed by the CRO and agreed upon with the sponsor before data base lock. (cf. DMP). For concomitant medications tables will show the frequencies of subjects by WHO DD preferred term.

### 5.6 Concomitant non-pharmacological measures, pre-medication

Not applicable.

### 5.7 PK and Efficacy

### 5.7.1 Pharmacokinetics

The primary objective of this study is the analysis of the PK profile of Wilate (refer to section 5.8).

### 5.7.2 Efficacy

All efficacy variables will be analyzed based on the FAS and additionally on the PP set, unless these analysis sets are identical.

Efficacy endpoints are:

- Efficacy of prophylactic treatment with *Wilate* based on the total annualized bleeding rate (TABR) as well as the spontaneous annualized bleeding rate (SABR)
- Efficacy of *Wilate* in the treatment of breakthrough BEs based on the proportion of BEs successfully treated with *Wilate* (successfully includes efficacy ratings assessed as either 'excellent' or 'good')
- Wilate consumption data (FVIII IU/kg per week and per month per subject) for prophylaxis



### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30

1100001101 712 0


Date of Issue: 2017-05-24


• Incremental IVR of *Wilate* over time (at baseline, and at 3 and 6 months of treatment) (refer to section 5.8)

### Efficacy of Prophylactic Treatment with Wilate

The analysis of the efficacy of prophylactic treatment with *Wilate* will be statistically evaluated by presenting descriptive sampling statistics for the TABR and SABR, along with an exploratory 95% CI for the mean. TABR and SABR will be calculated as the total number of BEs or total number of spontaneous BEs, respectively, in the time period between first dose of IMP and the study completion visit, divided by the duration (in years) between first dose of IMP and the study completion visit. Surgery periods, and BEs occurring within these periods, will be excluded from the calculation of annual bleeding rates

### Efficacy in the Treatment of Breakthrough BEs

To assess the hemostatic efficacy of *Wilate* in the treatment of breakthrough bleedings, a frequency distribution of all such BEs being successfully treated will be presented, along with an exploratory 95% CI.

Primarily, all obtained data on treatment characteristics (IMP dosages, frequencies, total consumption) and BEs (duration, frequency, efficacy assessment) will be described by providing summary statistics.

In general, the efficacy of bleeding episodes will also be presented by type (spontaneous, traumatic, postoperative, other), sites (nose, oral cavity, knee, ankle, elbow, arm, leg, intestinal and other. In addition, knee, ankle and elbow sites will be summarized as site 'joint') and severity (minor, moderate, major, life-threatening).

### Analysis of Other Secondary Endpoints

The statistical analysis of other secondary endpoints will be descriptive, including exploratory 95% CIs for the location parameters.

### 5.7.3 Exploratory Endpoint

An exploratory endpoint of this study is the descriptive efficacy of *Wilate* in surgical prophylaxis (for details see section 5.9).



|-----------------------------------------------|
| Date of Issue: 2017-05-24 |

### 5.8 Pharmacokinetics / Pharmacodynamics

For Pharmacokinetics and IVR assessments FVIII:C will be measured by both, the chromogenic (CHR) and one-stage assay (OS) and analyzed based on actual IMP potency (refer to section 8.1).

The PK profiles of *Wilate* and the PK parameters derived from them will be summarized by descriptive statistics as well as the presentation of concentration vs. time plots based on the PK set. In the analysis of the PK profiles geometric means and standard deviations will be presented in addition to the arithmetic means and standard deviations.

The following PK parameter will be derived and presented using a non-compartment model:

- Area under the curve (AUC) and AUC normalized for the administered dose (AUC<sub>norm</sub>)
- FVIII in vivo half-life  $(T_{1/2})$
- Maximum plasma concentration (C<sub>max</sub>)
- Time to reach maximum plasma concentration (T<sub>max</sub>)
- Mean residence time (MRT)
- Volume of distribution (Vd)
- Clearance (CL)
- Incremental in vivo recovery (IVR)

Analysis of variance (ANOVA) will be used in an exploratory sense to assess a possible association between AB0 blood type, VWF:Ag, and the FVIII:C half-life of *Wilate*.

Incremental IVR will be calculated from FVIII:C plasma levels measured before injection and peak levels obtained in the 15-min post-injection sample using actual IMP potencies. The results of the IVR assessments over time will be analyzed in summary tables for each time point and their differences to baseline along with 95% CIs for the mean differences.

### 5.9 Surgeries

Efficacy in surgical prophylaxis will be analyzed descriptively, presenting summary tables and listing on all aspects of surgical treatment and procedures as well as efficacy ratings.

The following surgery-related parameters will be presented:

- Number of minor and major surgeries
- Location, severity (minor or major, for definitions see protocol), and type (planned or emergency) of surgery
- Expected and actual duration of surgical procedure
- Expected and actual blood loss
- Pre-, intra-, and/or postoperative IMP administration data (only listed)




- Pre-, intra-, and postoperative FVIII plasma levels (only listed)
- VWF:Ag and VWF:Ac (descriptive statistics including changes to pre-infusion)
- Frequency and amount of blood transfusion requirements
- Presence of wound hematomas and whether or not they require surgical evacuation (only listed)
- Assessment of efficacy of surgical prophylaxis:
  - 1. at the end of surgery by the surgeon
  - 2. at end of the postoperative period by the hematologist
  - 3. Overall efficacy taking both the intra- and postoperative assessments into account assessed by the Investigator.
- Number of successively treated surgeries ('excellent' or 'good' overall efficacy rating)
- Concomitantly administered products (only listed)
- Narrative describing the outcome and efficacy of the intervention (only listed)
- Inhibitor testing (within 3–8 weeks after the end of the surgery, this visit may coincide with another study visit with scheduled inhibitor testing)

### 5.10 Safety

All safety analyses will be based on the SAF population.

The analysis of safety will include the occurrence of AEs, the results of the safety laboratory tests, immunogenicity measurements and the occurrence of parvovirus B19 seroconversions.

### 5.10.1 Adverse events

Adverse events (AEs) will be coded by the CRO according to the latest Medical Dictionary for Regulatory Activities (MedDRA). Coding will be agreed upon with the Sponsor before database lock (cf. DMP).

All adverse events recorded since signing of the informed consent form (ICF) will be listed in appendix 16.2 of the report differentiating by treatment emergent and non-treatment emergent events. This includes also post-study serious adverse events (SAEs) which occurred up to 4 weeks after the last IMP administration (not monitored proactively), thromboembolic events monitored proactively by performing a Follow-up Contact 30 days after the completion visit as well as safety relevant information on drug overdosing, drug interactions and medication errors.

The analysis will include only treatment-emergent adverse events (TEAEs), i.e. all documented AEs that started or worsened after the start of IMP infusion. It is assumed that for each increase in intensity of an AE a new entry of the AE will be done by the investigator; hence such cases will be analyzed like different phases of the same AE.



### Version Number: 1.1 Date of Issue: 2017-05-24 STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 

A descriptive analysis will be performed. Incidences will be presented by primary system organ classes (SOC) and incidences of PT within primary SOC sorted according to the Internationally Agreed Order.

Multiple counts within a PT or SOC (repeated or different included terms or changes in descriptors) will be counted only once for the calculation of incidences.

Global incidences will be calculated for:

- All TEAE irrespective of the causality assessment
- Related TEAEs ('Probably' or 'Possible')
- TEAEs by worst severity
- Serious TEAEs

A listing of "special cases" containing subject identification, age, sex, AE descriptors, start and end of treatment will be prepared for the following types of TEAEs:

- Serious adverse events (SAE)
- Adverse events which led to death
- Adverse events which led to discontinuation

Serious non-treatment emergent AEs will be listed separately.

### 5.10.2 Vital signs

Vital signs parameters (systolic/diastolic blood pressure, pulse, body weight, respiratory rates, body temperature) will be assessed at screening, PK visit, after 3 months at study completion visits and during surgery.

Descriptive analyses of values will be performed and changes from baseline will be analyzed for vital signs parameters at visits.

### 5.10.3 Safety laboratory variables

The analysis of the safety parameters (lab values for Hematology and Clinical chemistry) recorded during visits (screening, PK visit, 3-month and study completion visits) and at surgery will be purely descriptive and presented as summary tables or listings.

Time profiles of the safety laboratory parameters will be analyzed by presenting sampling statistics for the values as well as their difference to baseline at each time point. Additionally, frequency tables for values outside the normal ranges will be presented.

Similarly, time profiles of FVIII inhibitor testing results will be analyzed by presenting sampling statistics for the values as well as frequency tables for positive findings, along with 95% Pearson-Clopper CIs.




The thromboembolic risk will be monitored by determination of VWF:Ag and VWF:Ac during the study and especially postoperatively. Descriptive statistics including changes to preinfusion will be presented by visit and timepoint (with 95% CI) for visits or by operative day and timepoint for surgeries, respectively.

To assess the viral safety of *Wilate* incidences of parvovirus B19 seroconversions between baseline and end of study will be estimated along with 95% Pearson-Clopper CIs.

### 5.10.4 Other safety variables

Other safety parameters (e.g., changes in physical examination findings) will be analyzed by summary tables or listings. All abnormal findings from the physical examination will be listed.

The analysis of the safety parameters recorded during surgery (lab values) will be purely descriptive and presented as summary tables or listings.

### 5.11 Other variables

Not applicable.

### 5.12 Interim analyses

Not applicable.

### **6 QUALITY CONTROL**

The responsible project manager will review the SAP before it is provided to the Sponsor for review. The SAP will be signed off only when approval from the Sponsor's representative is received.

Log files of all SAS® programs needed for analysis will be checked for errors, warnings and suspicious notes by the statistical programmer. All findings will be either eliminated or commented upon. The final version of each program will be stored along with its log file in the electronic archive.

All programs will be validated by the author.

The agreement of the program outputs with the SAP, their consistency and plausibility will be checked by the TS. Moreover, the TS will review the outputs regarding completeness, readability and comprehensibility.

### **7 REFERENCES**

No specific references were used.



|-----------------------------------------------|--|


Date of Issue: 2017-05-24


### 8 APPENDICES

### 8.1 Formulas for derived variables

| Variable | Description |
|---|---|
| Actual potency | Potency of IMP (IU) based on central laboratory measurements of FVIII content by two assay methods: CHR (chromogenic) and OS (one-stage). |
| | The analysis of PK and IVR assessment will be based on actual potencies |
| Durations be-<br>tween two dates | Later date minus earlier date plus 1, expressed in days. (Remark: Duration will be 1, if both dates are the same.) |
| Annual bleeding rate | Number of bleeding / (last date of IMP – first date of IMP + 1)/365.25 |
| AUC | Area under the curve from baseline to infinity |
| | $AUC = \sum \left( \frac{(C_n + C_{n+1})}{2} \cdot \Delta t \right) + \frac{C_{last}}{K}$ |
| | ( $C_{last}$ is the last available measurement) |
| AUC <sub>norm</sub> | AUC normalized for the administered dose |
| AUMC | Area under the moment curve (from baseline to infinity) |
| | $AUMC = \sum \left( \frac{(t_n \cdot C_n + t_{n+1}C_{n+1})}{2} \cdot \Delta t \right) + \frac{C_{last}}{K^2} + \frac{t_{last} \cdot C_{last}}{K}$ |
| CL | Clearance |
| | $CL = \frac{D}{AUC}$ |
| | where $D$ is the actual dose administered (see remark above) |
| $C_0$ | FVIII concentration before IPM administration |
| C <sub>max</sub> | Maximal measured concentration after end of IMP infusion (peak concentration) |
| ED | Exposure day = each calendar day the subject received IMP |
| Incremental recovery (IVR) | $IVR = \frac{(C_{\text{max}} - C_0) \cdot BW}{D}$ |
| | where BW stands for the body weight in kg and D is the dose according to the actual potency of the FVIII concentrate as described in above |
| Labelled potency | Potency of IMP (IU) based on label of vial (IU). |




Date of Issue: 2017-05-24


| | Dosing analyses will be based on labelled potency |
|---|---|
| MRT | Mean residence time |
| | $MRT = \frac{AUMC}{AUC}$ |
| Success (for | Excellent or good efficacy rating |
| bleeding epi- | |
| sodes and sur- | |
| geries) | |
| $T_{1/2}$ | In vivo half-life |
| | using linear regression on the terminal phase of the logarithm of the concentration; |
| | $T_{\frac{1}{2}} = \frac{\ln(2)}{K}$ |
| | (where <i>K</i> , the elimination rate constant, is determined as the slope of the regression line) |
| $T_{\text{max}}$ | Time to reach maximum plasma concentration (Timing starts at end of infusion) |
| Vd | Volume of distribution |
| | $Vd = CL \cdot MRT$ |




Date of Issue: 2017-05-24


### 8.2 Algorithm for the Overall Efficacy Assessment for Surgical Prophylaxis

The evaluation of overall efficacy of the treatment in surgeries based on the intraoperative and postoperative assessment is defined as described below:

| Intraoperative | Postoperative assessment | | | |
|---|---|---|---|---|
| assessment | Excellent Good | | Moderate | None |
| Excellent | Excellent | Good | Good | Moderate |
| Good | Good | Good | Moderate | Moderate |
| Moderate | Good | Moderate | Moderate | None |
| None | Good | Moderate | None | None |




Date of Issue: 2017-05-24


### 8.3 List of Tables, Listings, Figures

A complete lists of tables, listings figures (TLFs) will be given in a separate document which can be updated without updating the SAP. The list will serve as a reference for both the Sponsor, the trial statistician and the statistical programmer and includes the totality of statistical output to be produced. Therefore, this list will be approved by both parties before commencing the statistical programming.

All output will be headed with an appropriate heading specifying the study ID and abbreviated study title.

All output will be dated and have page numbers in the form 'Page [x / y]' where x denotes the current page within an output and y the total number of pages of that output.

All statistical output will identify the underlying analysis populations and indicate the number of subjects / events in this population (N) and the number of subject/events actually contributing to the particular output (n). All statistical output will be presented per treatment group and in total (if applicable).

All subject listings will contain additionally to the subject identification the analysis population and the treatment group.




Version Number: 1.2

Date of Issue: 2019-07-08


| Sponsor: | Octapharma AG |
|---|---|
| Title of Protocol: | Clinical Study to Investigate the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of <i>Wilate</i> in Previously Treated Pediatric Patients with Severe Hemophilia A |
| Protocol Version/Date: | Version 02, 2017-06-19 (Ukraine only)<br>Version 03, 2018-07-06 |
| CRF Version: | Version 2.0, 2017-08-14 |
| Supersedes SAP Version: | Version 1.1, 2017-05-24 |


This document contains confidential information which must not be disclosed to anyone other than the involved CRO. This information should not be used for any purpose other than the evaluation of the clinical investigation without prior written consent of Octapharma.

No part of this document may be reproduced or stored in a retrieval system or transmitted in any other form or by any other means.




Date of Issue: 2019-07-08


### **Document authorization**



### **ERGOMED**

### STATISTICAL ANALYSIS PLAN


Date of Issue: 2019-07-08






### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.2 Date of Issue: 2019-07-08 

### Change control

| Date | Author | Reason | Version |
|---|---|---|---|
| 2017-04-26 | | | 1.0 |
| 2017-05-24 | | SAP adapted to protocol version 01, 15-May-2017 | 1.1 |
| 2019-07-08 | | Subgroup for bleeding analysis added as agreed at Database Review Meeting, formulas for derivations added | 1.2 |




Date of Issue: 2019-07-08


### TABLE OF CONTENTS

| Document authorization | |
|---|---|
| Consistency check with the Protocol (one option to be selected) | 3 |
| Change control | |
| Table of contents | |
| List of abbreviations | |
| 1 Study material | |
| 2 Study information | |
| 2.1 Primary objective | |
| 2.2 Secondary objective | |
| 2.3 Additional Objective: | |
| 2.4 Study design | |
| 2.5 Planned sample size | |
| 3 General Information | |
| 3.1 Background details | |
| 3.2 Deviations from the trial protocol with regard to statistical analyses | |
| 3.3 Individual protocol deviations | |
| 4 Analysis Populations | |
| 4.1 Safety set | |
| 4.2 Full analysis set | |
| 4.3 Pharmacokinetic set | |
| 4.4 Per-protocol set | |
| 4.5 Surgery set | |
| 4.6 Subgroup analyses | 15 |
| 5 Statistical Analyses | 15 |
| 5.1 Conventions | |
| 5.1.1 Baseline definition | |
| 5.1.2 Missing data | |
| 5.1.3 Pooling of centers | |
| 5.2 Demographic and other background data | |
| 5.2.1 Basic description | |
| 5.3 IMP exposure, compliance | |
| 5.4 Medical history | |
| 5.5 Concomitant medication | |
| 5.6 Concomitant non-pharmacological measures, pre-medication | |
| 5.7 PK and Efficacy | 18 |
| 5.7.2 Efficacy | |
| 5.7.3 Exploratory Endpoint | |
| 5.8 Pharmacokinetics / Pharmacodynamics | |
| 5.9 Surgeries | |
| 5.10 Safety | |
| 5.10.1 Adverse events | |
| 5.10.2 Vital signs | 22 |
| 5.10.3 Safety laboratory variables | |
| 5.10.4 Other safety variables | |
| 5.11 Other variables | |
| 5.12 Interim analyses | |
| 6 Quality Control | 23 |
| 7 References | |
| 8 Appendices | 24 |



# STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.2 Date of Issue: 2019-07-08 

| 8.1 | Formulas for derived variables | 24 |
|---|---|---|
| 8.2 | Algorithm for the Overall Efficacy Assessment for Surgical Prophylaxis | 26 |
| | List of Tables, Listings, Figures | |




Date of Issue: 2019-07-08


### LIST OF ABBREVIATIONS

Abbreviation Description

ABR Annual Bleeding Rate

AE Adverse Event

ANOVA Analysis of Variance
AUC Area Under the Curve

AUC normalized for the administered dose

AUMC Area Under the Moment Curve

BE Bleeding Episode
BMI Body Mass Index

BW Body Weight

CD4 Cluster of Differentiation 4

CHR Chromogenic assay
CI Confidence Interval

CL Clearance

C<sub>max</sub> Maximum Plasma Concentration

CRF Case Report Form

CRO Contract Research Organization

CSR Clinical Study Report

DD Drug Dictionary (WHO Coding Thesaurus)

DBR Database Review

DMP Data Management Plan

DVP Data Validation Plan

ED Exposure Day

EDC Electronic Data Capture

EOT End of Trial

eCRF Electronic Case Report Form

FAS Full Analysis Set

FVIII Coagulation Factor VIII

FVIII:C Factor VIII-coagulant




Date of Issue: 2019-07-08


Abbreviation Description

HJHS Hemophilia Joint Health Score

ICF Informed Consent Form

ID Identifier

IMP Investigational Medicinal Product

IRB Institutional Review Board

ITT Intention-To-Treat
IU International Unit

IV Intravenous

IVR Incremental in Vivo Recovery

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

MRT Mean Residence Time

N Number of Subjects/Observations

OS One-stage assay
PK Pharmacokinetic
POP Postoperative
PP Per-Protocol
PT Preferred Term

PTP Previously Treated Subject

QC Quality Control

SAE Serious Adverse Event

SAF Safety Analysis Set

SAP Statistical Analysis Plan

SAS Statistical Analysis Software package

SD Standard Deviation SOC System Organ Class

SOP Standard Operating Procedure

SABR Spontaneous Annualized Bleeding Rate

SURG Surgery analysis set




Date of Issue: 2019-07-08


| Abbreviation | Description |
|--------------|-------------------|
| $T_{1/2}$ | In Vivo Half-Life |
| TADD | 7T' ( 1 A 1'. 11 |

TABR Total Annualized Bleeding Rate

TEAE Treatment Emergent Adverse Event

TLFs Tables, Listings, Figures

T<sub>max</sub> Time to Reach Maximum Plasma Concentration

TS Trial Statistician

Vd Volume of distribution

VWD Von Willebrand Disease

VWF Von Willebrand Factor

VWF:Ac VWF activity

VWF:Ag Von Willebrand Factor Antigen

WHO World Health Organization



|-----------------------------------------------|---------------|
| Version Number: 1.2 | D 10 - 527 |
| Date of Issue: 2019-07-08 | |

### 1 STUDY MATERIAL

The following material was considered for this SAP:

| Document | Version, Date |
|----------|-------------------------|
| Protocol | Version 1.0, 2017-04-26 |
| CRF | TBD |
| DMP | TBD |
| DVP | TBD |
| DVP | TBD |

### 2 STUDY INFORMATION

### 2.1 Primary objective

The primary objective of this study is to determine the FVIII:C pharmacokinetics (PK) for *Wilate* in previously treated patients (PTP) with severe hemophilia A aged 1 to <12 years.

### 2.2 Secondary objective

The secondary objectives of this study are to:

- Determine the efficacy of *Wilate* in prophylactic treatment
- Determine the efficacy of *Wilate* in the treatment of breakthrough bleeding episodes (BEs)
- Calculate the FVIII:C incremental IVR of *Wilate* over time (at baseline, and at 3 and 6 months of treatment)
- Assess the association between AB0 blood type and the FVIII:C half-life of Wilate
- Assess the association between the VWF:Ag concentration and the FVIII:C half-life of *Wilate*
- Assess the safety and tolerability of Wilate
- Assess the immunogenicity of Wilate

### 2.3 Additional Objective:

An additional objective of this study is the descriptive efficacy of Wilate in surgical prophylaxis.




Date of Issue: 2019-07-08


### 2.4 Study design

This study is designed as a prospective, non-controlled, international, multi-center phase 3 study. Further details are given in the overview below:

### FLOW CHART FOR PK ASSESSMENT AND PROPHYLACTIC TREATMENT

| | Screen | PK<br>Visit | Pro<br>(starts wi | Follow-up<br>Contact<br>30 (±3) days<br>after | | | |
|---|---|---|---|---|---|---|---|
| | ing<br>Visit | | Day-14<br>Visit<br>(14–21<br>days) | Day-30<br>Visit<br>(±3<br>days) | 3-Month<br>Visit<br>(±2<br>weeks) | Study<br>Completion<br>(6-Month)<br>Visit<br>at 6 months<br>(+2 weeks) | Study Com-<br>pletion<br>Visit |
| Informed consent | Х | | | | | | |
| Inclusion and exclusion criteria | Х | | | | | | |
| Demographics | Х | | | | | | |
| Weight | Х | x [1] | | | x [1] | x [1] | |
| Height | Х | | | | | | |
| Medical history (incl. FVIII treatment 6 months before screening) | х | | | | | | |
| Vital signs | х | x [2] | | | x [4] | x [4] | |
| Physical examination | Х | | | | | х | |
| Routine safety laboratory | Х | x [3] | | | x [1] | x [4] | |
| Determination of CD4+ levels [8] | Х | | | | | | |
| Determination of AB0 blood group [9] | Х | | | | | | |
| HJHS, unless obtained within 3 months be-<br>fore screening | х | | | | | | |
| PK injection (50 ± 5 IU/kg) | | Х | | | | | |
| Blood sampling for FVIII:C (OS and CHR) for PK assessment | | x [5] | | | | | |
| IVR injection | | | | | Х | х | |
| Blood sampling for FVIII:C IVR (OS and CHR) | | | | | x [6] | x [6] | |
| Factor VIII inhibitor [10] | Х | x [1] | x [1] | x [1] | x [1] | x [1] | |
| VWF:Ag and VWF:Ac | | x [6] | x [1] | x [1] | x [6] | x [6] | |
| Parvovirus B19 antibodies | | x [1] | | | | x [7] | |
| Retention sample for possible virus marker testing | | x [1] | | | | | |
| Patient diary review | | | Х | Х | Х | х | |
| Adverse event monitoring | | Х | <b>»</b> | » | » | х | x [11] |
| Concomitant medications | Х | <b>»</b> | <b>»</b> | <b>»</b> | <b>»</b> | х | |

PK = pharmacokinetic, IVR = in vivo recovery, HJHS = Hemophilia Joint Health Score, OS = one-stage assay, CHR = chromogenic assay, VWF:Ag = von Willebrand factor antigen, VWF:Ac = VWF activity




Date of Issue: 2019-07-08


### LEGEND TO THE FLOW CHART FOR PK ASSESSMENT AND PROPHYLACTIC TREATMENT

- [1] Before injection
- [2] Before injection as well as 1 h (±5 min) and 48±2 h after injection
- [3] Before injection as well as 48±2 h after injection [local laboratory]
- [4] Before injection as well as 15±5 min after injection
- [5] Blood sampling within 1 h before injection and 15±5 min, 1 h (±5 min), 6 h (±30 min), 9±1 h, 24±2 h, and 48±2 h after the end of injection [central laboratory]
- [6] Blood sampling within 1 h before injection as well as 15±5 min after the end of injection [central laboratory]
- [7] If first sample was negative for parvovirus B19 antibodies (sample to be taken before injection) [central laboratory]
- [8] CD4+ count to be repeated if interval between Screening Visit and first injection exceeds 30 days. To be included into the study, the patient's CD4+ count must be >200/μL (i.e., inclusion criterion no. 4).
- [9] Unless obtainable from patient's medical history
- [10] Blood sampling for inhibitor testing should preferably be done at the time of trough FVIII:C levels [central laboratory]
  In case of positive inhibitor results, inhibitor retesting using a second, separately drawn sample should be performed, preferably within 15 days of becoming aware of the positive result.
- [11] Documentation of any thromboembolic events only (to be documented on AE page)




Date of Issue: 2019-07-08


### FLOW CHART OF ASSESSMENTS FOR SURGICAL PROPHYLAXIS

| | Within | Within | Surg | ery | POP<br>day 1 | Any<br>POP<br>day | End of<br>POP<br>period | 3-8<br>weeks<br>after<br>surgery |
|---|---|---|---|---|---|---|---|---|
| | 12 hours 3 hour before before | 3 hours<br>before<br>start | Intra-<br>opera-<br>tively | End<br>[1] | | | | |
| Body weight | х | | | | | | | |
| Type of surgery | Х | | | | | | | |
| Location of surgery | Х | | | | | | | |
| Severity of surgery | х | | | | | | | |
| Expected duration of surgery | Х | | | | | | | |
| Expected average/ maximum blood loss during surgery | Х | | | | | | | |
| Actual duration of surgery | | | | Х | | | | |
| Actual blood loss during surgery | | | | Х | | | | |
| Administration of IMP | | Х | (x) | (x) | (x) | (x) | (x) | |
| FVIII plasma levels | | # | (#) | (#) | # [2] | # | # | |
| VWF:Ag and VWF:Ac | | # | | | # [2] | # | # | |
| Presence of wound hematomas | | | | | х | х | х | |
| Routine safety laboratory | х | | | | (x) | (x) | (x) | |
| Vital signs | х | | Х | | х | | | |
| Efficacy assessment | | | | S | | | Н | |
| Overall efficacy assessment | | | | | | | ı | |
| Factor VIII inhibitor [3] | | | - | | | | | Х |
| Narrative of outcome | X | | | | | | | |
| Concomitant medications | throughout observation period | | | | | | | |
| Adverse event monitoring | throughout observation period | | | | | | | |

POP = postoperative, VWF:Ag = von Willebrand factor antigen, VWF:Ac = VWF activity

### 2.5 Planned sample size

Overall, 10 PTPs (5 patients aged 1 to <6 years of age and 5 patients aged 6 to <12 years) will be enrolled into this study. The aim is to obtain evaluable data on 8 patients who complete both the 2-day PK Phase and the 6-month Prophylactic Treatment Phase. Of the 8 evaluable patients, 4 patients must be 1 to <6 years of age, and another 4 patients must be 6 to <12 years of age. Enrolled patients will be replaced only if they do not complete the PK assessment.

The sample size of 10 pediatric patients to be enrolled was based on medical and regulatory reasoning. No statistical sample size estimation was performed.

<sup>()</sup> Optional

<sup>#</sup> Samples to be taken immediately before (≤ 30 min) and 30±15 min after IMP administration

<sup>[1]</sup> Time immediately after the last surgical suture

<sup>[2]</sup> For major surgeries, mandatory for the first 3 postoperative doses

<sup>[3]</sup> In case of positive inhibitor results, inhibitor retesting using a second, separately drawn sample should be performed, preferably within 15 days of becoming aware of the positive result.

S, performed by surgeon; H, performed by hematologist; I performed by Investigator



|---|---|---|
| Version Number | r: 1.2 | D14-527 |
| Date of Issue: | 2019-07-08 | |

### **3 GENERAL INFORMATION**

### 3.1 Background details

The data will be transferred to SAS from the Clinical Data Management System OPVERDI via a validated procedure. If applicable, external data will also be transferred to SAS for presentation of these data in the statistical analyses.

### 3.2 Deviations from the trial protocol with regard to statistical analyses

No deviations from the protocol are planned.

### 3.3 Individual protocol deviations

Any deviation from protocol will be discussed case by case before database lock whether the deviation has to be regarded as minor or as major (and therefore will lead to exclusion from particular analysis populations).

Examples for minor protocol violations may be deviations from scheduled investigation time.

Criteria for major protocol violations will at least include:

- Any substantial violation of in- or exclusion criteria.
- Use of concomitant medication that may interfere with the assessment of efficacy.

The final decision about the classification of individual protocol deviations and their consequences regarding assignment of subjects to analysis sets will be made during the data review meeting (DBR). A complete listing of protocol deviations and the judgment for assessment of subject disposition will be approved by the Sponsor and signed before database lock. All deviations along with the disposition of each subject will be recorded in a separate database member that will become part of the study database. A description of all major protocol violations will be included in the table part of the CSR.

### **4 ANALYSIS POPULATIONS**

The disposition of subjects will be displayed according to the following analysis populations:

- Safety (SAF) set
- Full Analysis set (FAS)
- Pharmacokinetic (PK) set
- Per-Protocol (PP) set
- Surgery (SURG) set




### 4.1 Safety set

The safety (SAF) set will include all subjects who received at least one infusion of IMP.

### 4.2 Full analysis set

The **full analysis set (FAS)** defined according to the intention-to-treat (ITT) principle will include all enrolled subjects who received at least one infusion of IMP (after the initial PK visit).

### 4.3 Pharmacokinetic set

The **pharmacokinetic (PK) set** will include all patients for which a valid *Wilate* PK profile has been obtained.

### 4.4 Per-protocol set

The **per-protocol (PP) set**, i.e. a subset of the FAS, will exclude subjects with major protocol deviations which may have an impact on the evaluation of the primary study outcome parameter (major protocol deviations as defined during DBR).

### 4.5 Surgery set

The **surgery (SURG) set** will be a subset of the FAS, containing all subjects who underwent a surgical procedure treated with *Wilate* during their Prophylactic Treatment Phase.

### 4.6 Subgroup analyses

The analyses of the PK parameters and the efficacy endpoints 'efficacy of prophylactic treatment' and 'efficacy in treatment of breakthrough BEs' will be presented by age groups ('1 to <6 years' and '6 to <12 years').

Efficacy analysis of secondary endpoint "efficacy of *Wilate* in the treatment of breakthrough (BEs) will be stratified by the following subgroups:

- Treatment-emergent bleeding episodes treated according to protocol ('BLEEDPP')
- Treatment-emergent bleeding episodes not treated according to protocol ('BLEED')

All bleeding events, which have not been treated with IMP or treatment significantly deviates from recommended treatment will be excluded from 'BLEED PP'.

Treatment with less than 25% of the lowest or more than 40% of the highest recommended dose in more than 50% of infusions administered for the corresponding event is considered as significant deviation.

### **5 STATISTICAL ANALYSES**

All statistical analyses will be performed using SAS® for Windows (Version 9.3 or later).

Descriptive statistics will always be given for the entire population.




The analysis of safety will be based on the SAF set.

Analysis of the PK properties of Wilate will be based on the PK set.

For secondary endpoints, FAS and PP analyses will be carried out, unless these analysis sets differ by no more than 1 patient from the FAS.

Analysis of the efficacy and safety of Wilate in surgeries will be based on the SURG set.

If not stated otherwise the following standard descriptive statistics will be presented:

### Descriptive statistics for continuous data

Number of subjects (N), arithmetic mean, standard deviation (SD), minimum, lower quartile, median, upper quartile and maximum will be presented. Usually mean and quartiles will have 1 decimal more, SD 2 decimals more than the original values (as given with min, max); N has no decimals. These descriptive statistics will be determined for measured values and for differences to baseline.

### Descriptive statistics for categorical data

Absolute frequencies (N) will be presented with 0, relative frequencies (%) with 1 decimal. For changes from baseline, shift tables may be generated.

### Inferential statistics

If not stated otherwise all statistical tests will be performed as described in the corresponding sections below.

All p-values will be rounded to 4 decimals (p<0.0001 will be displayed, if the p-values are less than 0.0001). Statistical significance will be declared if the rounded p-value will be less than 0.05.

All confidence intervals (CI) will be derived two-sided and at a confidence probability of 1- $\alpha = 0.95$ .

### Listings

All subject data will be listed by subject. Identification variable will be the subject ID (composed of study, center and subject number separated by a hyphen, e.g. '30-01-01'. Any derived data listed will also be stored permanently and will be calculated as outlined in section 8.1 of this SAP.

### 5.1 Conventions

### 5.1.1 Baseline definition

Assessments at PK visit or at screening visit (in case the corresponding assessment is not scheduled at PK visit) are considered as baseline.



|-----------------------------------------------|---------------|
| Version Number: 1.2 | Dags 17 of 27 |
| Date of Issue: 2019-07-08 | |

### 5.1.2 Missing data

In case of missing weight documentation data will be imputed using the Last Observation Carried Forward (LOCF) approach to calculate the dose per kg body weight (IU/kg). For calculation of PK parameters, missing measurements on a subject's PK profile will be handled according to the algorithms included in the PK software WinNonlin (version 7.0).

No further imputations for missing data will be performed.

Calculations pertaining to the derivation of annual bleeding rates will be based on documented time periods only.

### 5.1.3 Pooling of centers

All tables will be presented in total over all participating countries and centers. The distribution of number of subjects per country and center will be presented in the disposition section of the report.

### 5.2 Demographic and other background data

### 5.2.1 Basic description

The disposition of subjects (cf. Section 4) will be tabulated for the entire population. Details on protocol deviations will be listed.

Discontinued subjects will be described by frequency distributions including the reasons and in individual listings.

Demographic data (age, weight, height, BMI, race, ethnic group) will be summarized in tables and presented for the SAF and FAS population. Other baseline or background data, e.g. disease-specific information, will comprise descriptive tables for the SAF and FAS population for the following variables:

- Blood group
- Last CD4+ level before enrolment
- VWF:Ag, VWF:Ac levels at PK visit
- FVIII inhibitor level
- Vital Signs (Systolic and diastolic blood pressure, pulse and body temperature) at screening
- Physical examination (normal/abnormal) at screening
- Hemophilia joint health score (HJHS) at screening
- Results of Parvovirus B19 antibodies at PK visit

The following background data will only be listed:



# STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.2 Date of Issue: 2019-07-08 

• Medical history (including FVIII treatment during the last 6 months before screening)

Concomitant Medication

### 5.3 IMP exposure, compliance

Treatment will be administered prophylactically as defined in the protocol. Each home treatment will be recorded in the diary along with the reason for treatment (prophylaxis, bleeding, prevention of recurrent bleeding, prophylaxis after surgery or other reason). Treatments in context of IVR and PK measurements and surgeries will be documented in the patients notes. All treatments, from diary or patient's notes, will be transferred into the eCRF.

All IMP treatment details will be listed.

### 5.4 Medical history

Data on medical history will be listed. Medical history will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Codes will be reviewed by a Medical Expert and approved by the sponsor before data base lock.

### 5.5 Concomitant medication

Any relevant medication taken at time of screening and all new medications taken by the subject during the study period are defined as 'Concomitant'. Any changes of medications during the study period will also be recorded.

All details of concomitant medications will be listed including, the route, dose, frequency, start and stop date and indication.

Medications will be coded using the WHO DD thesaurus in the version current at the time of database lock. Coding will be performed by the CRO and agreed upon with the sponsor before data base lock. (cf. DMP). For concomitant medications tables will show the frequencies of subjects by WHO DD preferred term.

### 5.6 Concomitant non-pharmacological measures, pre-medication

Not applicable.

### 5.7 PK and Efficacy

### 5.7.1 Pharmacokinetics

The primary objective of this study is the analysis of the PK profile of Wilate (refer to section 5.8).




### 5.7.2 Efficacy

All efficacy variables will be analyzed based on the FAS and additionally on the PP set, unless these analysis sets are identical.

Efficacy endpoints are:

- Efficacy of prophylactic treatment with *Wilate* based on the total annualized bleeding rate (TABR) as well as the spontaneous annualized bleeding rate (SABR)
- Efficacy of *Wilate* in the treatment of breakthrough BEs based on the proportion of BEs successfully treated with *Wilate* (successfully includes efficacy ratings assessed as either 'excellent' or 'good')
- Wilate consumption data (FVIII IU/kg per week and per month per subject) for prophylaxis
- Incremental IVR of *Wilate* over time (at baseline, and at 3 and 6 months of treatment) (refer to section 5.8)

### Efficacy of Prophylactic Treatment with Wilate

The analysis of the efficacy of prophylactic treatment with *Wilate* will be statistically evaluated by presenting descriptive sampling statistics for the TABR and SABR, along with an exploratory 95% CI for the mean. TABR and SABR will be calculated as the total number of BEs or total number of spontaneous BEs, respectively, in the time period between first dose of IMP and the study completion visit, divided by the duration (in years) between first dose of IMP and the study completion visit. Surgery periods, and BEs occurring within these periods, will be excluded from the calculation of annual bleeding rates

### Efficacy in the Treatment of Breakthrough BEs

To assess the hemostatic efficacy of *Wilate* in the treatment of breakthrough bleedings, a frequency distribution of all such BEs being successfully treated will be presented, along with an exploratory 95% CI.

Primarily, all obtained data on treatment characteristics (IMP dosages, frequencies, total consumption) and BEs (duration, frequency, efficacy assessment) will be described by providing summary statistics.

In general, the efficacy of bleeding episodes will also be presented by type (spontaneous, traumatic, postoperative, other), sites (nose, oral cavity, knee, ankle, elbow, arm, leg, intestinal and other. In addition, knee, ankle and elbow sites will be summarized as site 'joint') and severity (minor, moderate, major, life-threatening).



|-----------------------------------------------|---------------|
| Version Number: 1.2 | Dago 20 of 27 |
| Date of Issue: 2019-07-08 | |

Analysis of Other Secondary Endpoints

The statistical analysis of other secondary endpoints will be descriptive, including exploratory 95% CIs for the location parameters.

### 5.7.3 Exploratory Endpoint

An exploratory endpoint of this study is the descriptive efficacy of <u>Wilate</u> in surgical prophylaxis (for details see section 5.9).

### 5.8 Pharmacokinetics / Pharmacodynamics

For Pharmacokinetics and IVR assessments FVIII:C will be measured by both, the chromogenic (CHR) and one-stage assay (OS) and analyzed based on actual IMP potency (refer to section 8.1).

The PK profiles of *Wilate* and the PK parameters derived from them will be summarized by descriptive statistics as well as the presentation of concentration vs. time plots based on the PK set. In the analysis of the PK profiles geometric means and standard deviations will be presented in addition to the arithmetic means and standard deviations.

The following PK parameter will be derived and presented using a non-compartment model:

- Area under the curve (AUC) and AUC normalized for the administered dose (AUC<sub>norm</sub>)
- FVIII in vivo half-life  $(T_{1/2})$
- Maximum plasma concentration (C<sub>max</sub>)
- Time to reach maximum plasma concentration (T<sub>max</sub>)
- Mean residence time (MRT)
- Volume of distribution (Vd)
- Clearance (CL)
- Incremental in vivo recovery (IVR)

Analysis of variance (ANOVA) will be used in an exploratory sense to assess a possible association between AB0 blood type, VWF:Ag, and the FVIII:C half-life of *Wilate*.

Incremental IVR will be calculated from FVIII:C plasma levels measured before injection and peak levels obtained in the 15-min post-injection sample using actual IMP potencies. The results of the IVR assessments over time will be analyzed in summary tables for each time point and their differences to baseline along with 95% CIs for the mean differences.

### 5.9 Surgeries

Efficacy in surgical prophylaxis will be analyzed descriptively, presenting summary tables and listing on all aspects of surgical treatment and procedures as well as efficacy ratings.



# STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.2 Date of Issue: 2019-07-08 

The following surgery-related parameters will be presented:

- Number of minor and major surgeries
- Location, severity (minor or major, for definitions see protocol), and type (planned or emergency) of surgery
- Expected and actual duration of surgical procedure
- Expected and actual blood loss
- Pre-, intra-, and/or postoperative IMP administration data (only listed)
- Pre-, intra-, and postoperative FVIII plasma levels (only listed)
- VWF:Ag and VWF:Ac (descriptive statistics including changes to pre-infusion)
- Frequency and amount of blood transfusion requirements
- Presence of wound hematomas and whether or not they require surgical evacuation (only listed)
- Assessment of efficacy of surgical prophylaxis:
  - 1. at the end of surgery by the surgeon
  - 2. at end of the postoperative period by the hematologist
  - 3. Overall efficacy taking both the intra- and postoperative assessments into account assessed by the Investigator.
- Number of successively treated surgeries ('excellent' or 'good' overall efficacy rating)
- Concomitantly administered products (only listed)
- Narrative describing the outcome and efficacy of the intervention (only listed)
- Inhibitor testing (within 3–8 weeks after the end of the surgery, this visit may coincide with another study visit with scheduled inhibitor testing)

### 5.10 Safety

All safety analyses will be based on the SAF population.

The analysis of safety will include the occurrence of AEs, the results of the safety laboratory tests, immunogenicity measurements and the occurrence of parvovirus B19 seroconversions.

### 5.10.1 Adverse events

Adverse events (AEs) will be coded by the CRO according to the latest Medical Dictionary for Regulatory Activities (MedDRA). Coding will be agreed upon with the Sponsor before database lock (cf. DMP).

All adverse events recorded since signing of the informed consent form (ICF) will be listed in appendix 16.2 of the report differentiating by treatment emergent and non-treatment emergent events. This includes also post-study serious adverse events (SAEs) which occurred up to 4



# STATISTICAL ANALYSIS PLAN Protocol No: WIL-30 Version Number: 1.2 Date of Issue: 2019-07-08 

weeks after the last IMP administration (not monitored proactively), thromboembolic events monitored proactively by performing a Follow-up Contact 30 days after the completion visit as well as safety relevant information on drug overdosing, drug interactions and medication errors.

The analysis will include only treatment-emergent adverse events (TEAEs), i.e. all documented AEs that started or worsened after the start of IMP infusion. It is assumed that for each increase in intensity of an AE a new entry of the AE will be done by the investigator; hence such cases will be analyzed like different phases of the same AE.

A descriptive analysis will be performed. Incidences will be presented by primary system organ classes (SOC) and incidences of PT within primary SOC sorted according to the Internationally Agreed Order.

Multiple counts within a PT or SOC (repeated or different included terms or changes in descriptors) will be counted only once for the calculation of incidences.

Global incidences will be calculated for:

- All TEAE irrespective of the causality assessment
- Related TEAEs ('Probably' or 'Possible')
- TEAEs by worst severity
- Serious TEAEs

A listing of "special cases" containing subject identification, age, sex, AE descriptors, start and end of treatment will be prepared for the following types of TEAEs:

- Serious adverse events (SAE)
- Adverse events which led to death
- Adverse events which led to discontinuation

Serious non-treatment emergent AEs will be listed separately.

### 5.10.2 Vital signs

Vital signs parameters (systolic/diastolic blood pressure, pulse, body weight, respiratory rates, body temperature) will be assessed at screening, PK visit, after 3 months at study completion visits and during surgery.

Descriptive analyses of values will be performed and changes from baseline will be analyzed for vital signs parameters at visits.




### 5.10.3 Safety laboratory variables

The analysis of the safety parameters (lab values for Hematology and Clinical chemistry) recorded during visits (screening, PK visit, 3-month and study completion visits) and at surgery will be purely descriptive and presented as summary tables or listings.

Time profiles of the safety laboratory parameters will be analyzed by presenting sampling statistics for the values as well as their difference to baseline at each time point. Additionally, frequency tables for values outside the normal ranges will be presented.

Similarly, time profiles of FVIII inhibitor testing results will be analyzed by presenting sampling statistics for the values as well as frequency tables for positive findings, along with 95% Pearson-Clopper CIs.

The thromboembolic risk will be monitored by determination of VWF:Ag and VWF:Ac during the study and especially postoperatively. Descriptive statistics including changes to preinfusion will be presented by visit and timepoint (with 95% CI) for visits or by operative day and timepoint for surgeries, respectively.

To assess the viral safety of *Wilate* incidences of parvovirus B19 seroconversions between baseline and end of study will be estimated along with 95% Pearson-Clopper CIs.

### 5.10.4 Other safety variables

Other safety parameters (e.g., changes in physical examination findings) will be analyzed by summary tables or listings. All abnormal findings from the physical examination will be listed.

The analysis of the safety parameters recorded during surgery (lab values) will be purely descriptive and presented as summary tables or listings.

### 5.11 Other variables

Not applicable.

### 5.12 Interim analyses

Not applicable.

### **6 QUALITY CONTROL**

The responsible project manager will review the SAP before it is provided to the Sponsor for review. The SAP will be signed off only when approval from the Sponsor's representative is received.



|-----------------------------------------------|----------|
| Version Number: 1.2 | D 24 627 |
| Date of Issue: 2019 | |

Log files of all SAS® programs needed for analysis will be checked for errors, warnings and suspicious notes by the statistical programmer. All findings will be either eliminated or commented upon. The final version of each program will be stored along with its log file in the electronic archive.

All programs will be validated by the author.

The agreement of the program outputs with the SAP, their consistency and plausibility will be checked by the TS. Moreover, the TS will review the outputs regarding completeness, readability and comprehensibility.

### 7 REFERENCES

No specific references were used.

### **8 APPENDICES**

### 8.1 Formulas for derived variables

| Variable | Description |
|---|---|
| Actual potency | Potency of IMP (IU) based on central laboratory measurements of FVIII content by two assay methods: CHR (chromogenic) and OS (one-stage). The analysis of PK and IVR assessment will be based on actual poten- |
| | cies |
| Durations be-<br>tween two dates | Later date minus earlier date plus 1, expressed in days. (Remark: Duration will be 1, if both dates are the same.) |
| Spontaneous annualized bleeding rate (SABR) | Number of spontaneous bleedings (excluding bleedings occurring in surgery periods) between first dose of IMP and Study Completion visit (or last dose of IMP in case completion visit not performed) / time under prophylaxis (days)/365.25 (see prophylactic treatment phase) |
| Total annualized<br>bleeding rate<br>(TABR) | Number of bleedings (excluding bleedings occurring in surgery periods) between first dose of IMP and Study Completion visit (or last dose of IMP in case completion visit not performed / time under prophylaxis (days)/365.25 (see prophylactic treatment phase) |
| Surgery Phase | Last treatment for surgery – first treatment for surgery + 1 |
| Prophylactic treatment phase | Date of completion visit or date of last treatment with IMP in case completion visit not performed) – (date of first prophylactic treatment after the PK visit) + 1 – Surgery phases |
| Time in study | Date of study completion – date of screening +1 |




Date of Issue: 2019-07-08


| Variable | Description |
|---|---|
| Time under treat- | Date of last treatment – date of first treatment + 1 (average drug con- |
| ment | sumption data will be calculated relative to time under treatment) |
| AUC | Area under the curve from baseline to infinity |
| | $AUC = \sum \left( \frac{(C_n + C_{n+1})}{2} \cdot \Delta t \right) + \frac{C_{last}}{K}$ |
| | ( $C_{last}$ is the last available measurement) |
| AUC <sub>norm</sub> | AUC normalized for the administered dose |
| AUMC | Area under the moment curve (from baseline to infinity) |
| | $AUMC = \sum \left( \frac{(t_n \cdot C_n + t_{n+1}C_{n+1})}{2} \cdot \Delta t \right) + \frac{C_{last}}{K^2} + \frac{t_{last} \cdot C_{last}}{K}$ |
| CL | Clearance |
| | $CL = \frac{D}{AUC}$ |
| | where $D$ is the actual dose administered (see remark above) |
| $C_0$ | FVIII concentration before IPM administration |
| C <sub>max</sub> | Maximal measured concentration after end of IMP infusion (peak concentration) |
| ED | Exposure day = each calendar day the subject received IMP |
| Incremental re-<br>covery (IVR) | $IVR = \frac{(C_{\text{max}} - C_0) \cdot BW}{D}$ |
| | where BW stands for the body weight in kg and D is the dose according to the actual potency of the FVIII concentrate as described in above |
| Labelled potency | Potency of IMP (IU) based on label of vial (IU). Dosing analyses will be based on labelled potency |
| MRT | Mean residence time |
| | $MRT = \frac{AUMC}{AUC}$ |
| Success (for<br>bleeding epi-<br>sodes and sur-<br>geries) | Excellent or good efficacy rating |



|---|---|
| Version Number: 1 | Version Number: 1.2 |
| Date of Issue: 2 | |

| Variable | Description |
|---|---|
| $T_{1/2}$ | In vivo half-life |
| | using linear regression on the terminal phase of the logarithm of the concentration; |
| | $T_{\frac{1}{2}} = \frac{\ln(2)}{K}$ |
| | (where <i>K</i> , the elimination rate constant, is determined as the slope of the regression line) |
| $T_{\text{max}}$ | Time to reach maximum plasma concentration (Timing starts at end of infusion) |
| Vd | Volume of distribution |
| | $Vd = CL \cdot MRT$ |

### 8.2 Algorithm for the Overall Efficacy Assessment for Surgical Prophylaxis

The evaluation of overall efficacy of the treatment in surgeries based on the intraoperative and postoperative assessment is defined as described below:

| Intraoperative assessment | Postoperative assessment | | | |
|---|---|---|---|---|
| | Excellent | Good | Moderate | None |
| Excellent | Excellent | Good | Good | Moderate |
| Good | Good | Good | Moderate | Moderate |
| Moderate | Good | Moderate | Moderate | None |
| None | Good | Moderate | None | None |



### STATISTICAL ANALYSIS PLAN Protocol No: WIL-30


Date of Issue: 2019-07-08


### 8.3 List of Tables, Listings, Figures

A complete lists of tables, listings figures (TLFs) will be given in a separate document which can be updated without updating the SAP. The list will serve as a reference for both the Sponsor, the trial statistician and the statistical programmer and includes the totality of statistical output to be produced. Therefore, this list will be approved by both parties before commencing the statistical programming.

All output will be headed with an appropriate heading specifying the study ID and abbreviated study title.

All output will be dated and have page numbers in the form 'Page [x / y]' where x denotes the current page within an output and y the total number of pages of that output.

All statistical output will identify the underlying analysis populations and indicate the number of subjects / events in this population (N) and the number of subject/events actually contributing to the particular output (n). All statistical output will be presented per treatment group and in total (if applicable).

All subject listings will contain additionally to the subject identification the analysis population and the treatment group.